





**Cognitive Behavioral Analysis System of Psychotherapy (CBASP)** vs. Behavioral Activation (BA) in persistently depressed treatment-resistant inpatients: Efficacy, moderators, and mediators of change **Acronym: ChangePDD** 

NCT Number: NCT04996433

Document Date: 16.06.2021







University Greifswald
Clinical Psychology and Psychotherapy
Franz-Mehring Str. 47
17487 Greifswald

# **Study Protocol**

Cognitive Behavioral Analysis System of Psychotherapy (CBASP)
vs. Behavioral Activation (BA)
in persistently depressed treatment-resistant inpatients:
Efficacy, moderators, and mediators of change
Acronym: ChangePDD

Cognitive Behavioral Analysis System of Psychotherapy (CBASP) vs.
Behavioral Activation (BA) bei stationären Patienten mit persistierend depressiven und therapieresistenten Störungen:
Wirksamkeit, Moderatoren und Mediatoren der Veränderung

Version 3.0; 16.06.2021

### **Coordinating Investigator**

Prof. Dr. Eva-Lotta Brakemeier University Greifswald Clinical Psychology and Psychotherapy Franz-Mehring-Str. 47 17487 Greifswald

Email: <a href="mailto:eva-lotta.brakemeier@uni-greifswald.de">eva-lotta.brakemeier@uni-greifswald.de</a>
Phone.: +49 3834 420 3786 Fax: +49 3834 420 3736

# **Table of Contents**

| 1. | Study Synopsis | 7 |
|------|-------------------------------------------------|----|
| 2. | Responsibilities and Cooperation | 9 |
| 2.1. | . Responsibilities | 9 |
| 2.1. | .1. Investigator's responsibilities | 9 |
| 2.1. | .2. Further responsibilities | 10 |
| 2.2. | . Coordinating and Participating Sites | 10 |
| 2.3 | . Financial support | 12 |
| 2.4. | . Signature and Consent statement | 12 |
| 3. | Scientific Background | 19 |
| 4. | Rationale and Hypothesis | 20 |
| 4.1. | . Rationale | 20 |
| 4.2 | . Hypothesis | 21 |
| 5. | Study Design | 21 |
| 6. | Outcome Measures | 23 |
| 6.1 | . Primary Endpoint | 23 |
| 6.2 | . Secondary Endpoints, Moderators and Mediators | 24 |
| 6.3 | . Further Endpoints | 25 |
| 7. | Methods of Data collection | 26 |
| 8. | Study Population | 26 |
| 8.1. | . Treatment groups | 26 |
| 8.2. | . Inclusion criteria | 27 |
| 8.3 | . Exclusion criteria | 27 |
| 8.4 | . Methods against bias | 27 |
| 8.4 | .1. Randomization | 27 |
| 8.4 | .2. Blinding | 28 |
| 8.4 | .3. Control of therapy allegiance | 28 |
| 8.4 | .4. Control of overlapping treatments | 29 |
| 8.4 | .5. Control of confounding factors | 30 |
| 8.4 | .6. Control of measurement bias | 30 |
| 9. | Study Procedure | 30 |
| 9.1. | . Study visit overview | 30 |

| 9.2. \ | /isit 1 | 31 |
|---|---|---|
| 9.3. \ | /isit 2-5 | 32 |
| 9.4. \ | /isit 6-8 | 32 |
| 9.5. \ | /isit 9-11 | 32 |
| 9.6. \ | /isit 12-17 | 32 |
| 9.7. ( | Conduction of the Interventional Arm (CBASP) | 32 |
| 9.8. ( | Conduction of the Control Arm (BA) | 33 |
| 9.9. ( | Concomitant Therapy | 34 |
| 9.10. 9 | Study Sites | 36 |
| 9.11. ٦ | Freatment after end of study | 36 |
| 9.12. 9 | Study Schedule | 36 |
| 10. Ac | ld-on Studies | 37 |
| 10.1 C | hangePDD-EMA | 37 |
| 10.1.1 | Theoretical motivation | 37 |
| 10.1.1 | 2 ChangePDD-EMA study design | 38 |
| 10.1.2 | ChangePDD-EMA data assessment and analysis | 39 |
| 10.2 E | ffort Task | 40 |
| 10.2.1 | Theoretical motivation and hypotheses | 41 |
| 10.2.2 | Task and computational model | 41 |
| 10.2.3 | Study design | 42 |
| 10.3 S | tudy design and instruments supplemented by add-on studies | 43 |
| 11. Sa | fety | 44 |
| 11.1. <i>A</i> | Adverse reactions | 44 |
| 11.2. F | Risk-benefit-assessment | 45 |
| 11.2.1 | . Potential risks | 45 |
| 11.2.2 | . Potential benefit | 46 |
| 11.2.3 | . Conclusion | 46 |
| 11.3. [ | Discontinuation criteria | 47 |
| 11.3.1 | . Premature discontinuation of a patient | 47 |
| 11.3.2 | Premature discontinuation of the study | 47 |
| 11.4. [ | Data Monitoring Committee (DMC) | 48 |
| 12. Et | hical and regulatory aspects | 48 |
| 12.1. l | aws and regulations | 48 |
| 12.2. I | ndependent ethics committee | 48 |
| 12.3. ( | Changes to the study protocol | 48 |

| 12.4. Informed consent and insurance | 49 |
|-------------------------------------------------|----|
| 12.5. Data safety | 49 |
| 13. Statistics | 49 |
| 13.1. Sample size | 49 |
| 13.2. Statistical evaluation | 50 |
| 13.2.1. Primary endpoint | 50 |
| 13.2.2. Secondary endpoints | 51 |
| 13.2.3. Safety and tolerability endpoints | 51 |
| 13.2.4. Handling of dropouts | 51 |
| 14. Data Management | 51 |
| 14.1. Data collection | 51 |
| 14.2. Data processing | 52 |
| 13.2.1 EDC-System (eCRF) | 52 |
| 13.2.2 Data concealment for electronic transfer | 52 |
| 13.2.3 Data discrepancies | 52 |
| 13.2.4 Registration | 52 |
| 13.2.5 Publication | 53 |
| 13.2.6 Open Data | 53 |
| 14.3. Quality assurance and quality control | 53 |
| 14.3.1. Source data and subject files | 53 |
| 14.3.2. Monitoring | 54 |
| 15. Literature | 54 |

# List of Abbreviations

| Abbreviation | Definition |
|---|---|
| AE | Adverse Event |
| ATHF-SF | Antidepressant Treatment History Form - Short Form |
| ATR | Adverse Treatment Reaction |
| ВА | Behavioral Activation |
| BADS | Behavioral Activation Depression Scale |
| BDI-II | Beck's Depression Inventory |
| BDNF | Brain-Derived Neurotrophic Factor |
| BRS | Brief Resilience Scale |
| BSI | Brief Symptom Inventory |
| CBASP | Cognitive Behavioral Analysis System of Psychotherapy |
| CBASP-CAR /<br>BA-CAR | Observer based Competence and Adherence Rating of CBASP / BA |
| CBT | Cognitive Behavioral Therapy |
| CRF | Case Report Form |
| СТQ | Childhood Trauma Questionnaire |
| DAS | Dysfunctional Attitude Scale |
| DIPS | Diagnostic Interview for Mental Disorders |
| DMC | Data Monitoring Committee |
| DSM | Diagnostic and Statistical Manual of Mental Disorders |
| EC | Ethics Committee |
| ECR-RD8 | Experience in Close Relationships – Revised 8-item version |
| eCRF | Electronic Case Report Form |
| ECT | Electroconvulsive Therapy |
| EDC | Electronic Data Capture |
| ES | Euthymia Scale |
| FPFV | First Patient First Visit |
| GAF | Global Assessment of Functioning |
| GSE | General Self-Efficacy Scale |
| HDRS-24 | Hamilton Depression Rating Scale, 24-item version |

| Abbreviation Definition | |
|---|---|
| ICH-GCP | International Conference on Harmonization - Good Clinical Practice |
| IDS-SR | Inventory of Depressive Symptoms, Self-Report |
| IIP-32-R | Inventory of Interpersonal Problems, 32-item version, revised |
| IMI-R | Impact Message Inventory – Revised |
| ISF | Investigator Site File |
| ITT | Intention to Treat |
| KKS | Coordinating Center for Clinical Trials |
| LMM | Linear Mixed-effects Models |
| LQPT | Lübecker Questionnaire of Preoperational Thinking |
| LPLV | Last Patient Last Visit |
| MINI-ICF | Measure of disorders of capacity as defined by the International Classification of Function |
| MPQ | Mental Pain Questionnaire |
| PDD | Persistent Depressive Disorder |
| PI | Principal Investigator (Coordinating Investigator) |
| PID5BF + M | Personality Inventory for DSM-5 Brief Form Plus Modified |
| RCT | Randomized Controlled Trial |
| R-GPTS | Revised-Green Paranoid Thoughts Scale |
| RSQ | Rejection Sensitivity Questionnaire |
| SAB | Scientific Advisory Board |
| SAE | Severe Adverse Event |
| SATR | Severe Adverse Treatment Reaction |
| SCID-PD | Structured Clinical Interview for DSM-5 – Personality Disorders |
| SEPIPS | Side Effects of Psychological Interventions Process Scale |
| SNI | Social Network Index |
| TR | Treatment-Resistance |
| UCLA | UCLA Loneliness Scale |
| WAI | Working Alliance Inventory |
| WHO-5 | Well-Being Index |
| WHOQoL | World Health Organization Quality of Life |

# 1. Study Synopsis

| Title of the Study | Cognitive Behavioral Analysis System of Psychotherapy (CBASP) vs.<br>Behavioral Activation (BA) in persistently depressed treatment-<br>resistant inpatients: Efficacy, moderators, and mediators of change |
|---|---|
| Study Acronym | ChangePDD |
| Coordinating Investigator | Prof. Dr. Eva-Lotta Brakemeier |
| Indication | Persistent depressive disorder (PDD) with treatment-resistance (TR) |
| Objectives | To compare CBASP conducted over 16 weeks (acute and continuation treatment) with BA (same dose and duration) in PDD inpatients with TR regarding efficacy, moderators and mediators of change |
| Study Design | Prospective, multicenter, evaluator-blinded, parallel-group, randomized controlled intervention trial with an active control condition |
| Number of Patients | To be assessed for eligibility: n = 1000 to be screened at sites To be allocated to study: n = 396 To be analyzed: n = 396; Intention to Treat (ITT) Sample, 14% expected dropout included |
| Randomization | Randomization with stratification for severity of depression and study site with an allocation ratio of 1:1 |
| Eligibility Criteria - Inclusion | <ul> <li>Age 20-70 years</li> <li>Primary DSM-5 diagnosis of PDD (300.4, 296.2x, 296.3x)</li> <li>Total Hamilton Depression Rating Scale (HDRS-24) Score ≥ 20</li> <li>Treatment-resistance (TR) (defined as a level of 3 or higher on the ATHF-SF or medication intolerance or one psychotherapy at least 25 sessions by a certified therapist in the current episode)</li> <li>Sufficient knowledge of the German language</li> <li>Written informed consent</li> </ul> |
| Eligibility Criteria - Exclusion | <ul> <li>Bipolar I or II disorder</li> <li>Active substance use disorders (abstinence shorter than 6 months)</li> <li>Schizophrenia spectrum and other psychotic disorders</li> <li>Antisocial personality disorder</li> <li>Acute suicidality</li> <li>Previous CBASP or BA treatment within the last year</li> <li>Inability to tolerate CBASP or BA (e.g., organic brain disorders, severe cognitive deficits)</li> <li>Inability to participate in dayclinic or outpatient continuation treatment</li> </ul> |
| Test and Reference Treatment | Experimental intervention: CBASP Control intervention: BA |
| Time schedule | <ul> <li>Study treatment per patient: 112 days (16 weeks)</li> <li>Study duration per patient: 448 days (64 weeks, incl. follow-up)</li> <li>First patient first visit (FPFV) to last patient last visit (LPLV): 34 months (without follow-up), 46 months (incl. follow-up)</li> <li>Duration of the entire study: 58 months</li> <li>Recruitment period: 30 months</li> </ul> |

| Primary endpoint | Change in depression severity (HDRS-24 score) after 16 weeks |
|---|---|
| Secondary and further endpoints | Secondary endpoints: Depressive and anxiety symptomatology (HDRS-24 and IDS-SR) assessed every second week during treatment and at week 64; IDS-SR also measured every second month during follow-up Specific other important psychological variables (BSI, GAF, WHOQoL) assessed at week pre, 1, 5, 10, 16, and 64 Response, remission, dropout and relapse rates (according to HRSD-24 and hospitalization rates) assessed at week 5, 10, 16 and 64 (relapse rate only at week 16 and 64) costs and benefits (cost interview) assessed at week pre, 16, 64 Further endpoints: Other interesting psychological variables (BDI-II, BRS, DAS, ECR-D(, ES, IMI-R, LQPT, Mini-ICF, MPQ, PID5BF+M, R-GPTS, RSQ, SES, SNI, UCLA, WBI, WHOQOL, WHO-5) assessed at week pre, 1, 5, 10, 16, and 64 Main moderators (assessed at baseline): Childhood maltreatment (CTQ) Epigenetic (BDNF methylation) Main mediators (assessed at baseline and week 1, 2, 4, 6, 8, 10, 12, 14, 16, and 64): Interpersonal problems (IIP-32-R) Activities (BADS, actimeter-measured step-counts) Mediators only included in the two add-on studies: Interpersonal Activation Diary (IAD; assessed daily at week 0, 1, 2, 3, 4, 5, 6) Social interaction and current mood (assessed daily at week 0, 6) Effort Task (assessed at week 1, 5, 16) Safety: (Severe) Adverse events, negative effects including side effects (SEPIPS) and medication will be monitored |
| Statistical analysis | Description of the primary efficacy analysis and population: (Generalized) Linear Mixed-effects Models (LMM) with random intercepts and slopes predicting outcomes from time, treatment group, and time x treatment group interaction based on the Intention to Treat (ITT) sample Secondary endpoints Sensitivity analyses: - LMMs with covariates - LMMs based on the completer sample - Pattern-mixture Models Moderator analyses: - LMMs with covariate x time x group interactions Mediator analyses: - Dynamic Panel Models |
| Participating sites | No. of sites to be involved: six 1) Berlin, Charité, University Medicine Berlin 2) Hannover, Hannover Medical School 3) Lübeck, University Hospital of Lübeck 4) Marburg, University Hospital of Marburg 5) München, University Hospital of München 6) Tübingen, University Hospital of Tübingen |

# 2. Responsibilities and Cooperation

### 2.1. Responsibilities

The following Figure 1 gives an overview of all persons, committees, boards and sites involved in the study ChangePDD.



Figure 1: Persons, committees, boards and sites involved in the study ChangePDD

#### 2.1.1. Investigator's responsibilities

The **Principal Investigator (PI)** / **Coordinating Investigator (CI)** Prof. Dr. Eva-Lotta Brakemeier is a highly experienced scientist and psychotherapist and has sufficient experience in conducting clinical studies. She is responsible for the project coordination and project management, especially for conducting the clinical study in accordance with this study protocol, the ethical principles that have their origin in the Declaration of Helsinki (current version) as well as with ICH Guideline for Good Clinical Practice (ICH-E6 (R2)) and the relevant national laws and applicable regulatory requirements.

In particular, during the whole trial, she will keep the regular contact to all study parties for clinical and organizational questions including regular newsletters. For the initiation, she has to review and design the study protocol, study manuals, patient information, and informed consent form; in addition, she will revise the eCRF and coordinate the training of the participating sites and therapists as well as provide working instructions. During the

recruitment phase, she is responsible to revise the study documents, schedule the investigator meetings and presentations, participate in the meetings with project management at KKS, coordinate the training and supervision, communicate with and participate on meetings with DMC, progress reporting, generation and review of amendments, as well as supervise and evaluate SAE reports. During the follow up phase, she will coordinate the CBASP- and BA-CAR ratings as quality assurance and start preparation of the final reports. Concerning the analysis, she will prepare the final reports, presentations, and publications.

She is supported in all these tasks by Maike Hollandt, the **Clinical Project Management**, and Dr. Tim Kaiser, an expert in psychotherapy research, located at the University of Greifswald.

### 2.1.2. Further responsibilities

To successfully manage the trial, the KKS Greifswald, the Trial Steering Committee and the six Participating Sites will cooperate intensively while being supported by the DMC and the SAB (see Fig. 1).

The KKS Greifswald will support and mainly perform the study coordination. The KKS Greifswald is responsible for support concerning preparing and review of the clinical trial protocol and the informed consent form as well as the application to the ethics committees. Furthermore, the eCRF system will be managed by the KKS Greifswald. Monitoring will also be provided.

The **Statistician** Prof. Dr. Johannes Zimmermann is responsible for biometrics. In the initiation phase, he draws up the statistical analysis plan as well as standards for the data management and conceptualizes the eCRF and specific data formats. In the recruitment and follow-up phase, he prepares safety analyses and reports these to the DMC. The main task is the blinded analysis of the data and the provision of the final statistical analysis. In all these tasks, he is supported by a coworker at pre- or post-doc level.

The **Leading Investigators** of each site are responsible for recruiting and conducting study treatments while the **Core Scientists** support recruitment and conduction of study treatments as well as trainings and supervision.

Further responsibilities will be specified in separate contracts between the participating parties.

### 2.2. Coordinating and Participating Sites

Table 1 lists all six participating sites including the respective leading investigators and core scientists (main contact persons) as well as the addresses.

**Table 1:** Six participating clinical sites including the respective leading investigators and core scientists (main contact persons)

#### Charité, Universitätsmedizin Berlin

Klinik für Psychiatrie und Psychotherapie (CCM)

Charité - Universitätsmedizin Berlin

Charitéplatz 1 10117 Berlin

Prof. Dr. Philipp Sterzer (<a href="mailto:philipp.sterzer@charite.de">philipp.sterzer@charite.de</a>)

Tel.: +49-30-450-517215 / Fax: +49-30-450-517944 Prof. Dr. Stephan Köhler (stephan.koehler@charite.de)

Tel.: +49-30-450-617405 / Fax: +49-30-450-517903

#### Medizinische Hochschule Hannover

Klinik für Psychiatrie, Sozialpsychiatrie und Psychotherapie

Medizinische Hochschule Hannover

Carl-Neuberg-Straße 1

30625 Hannover

Prof. Dr. Kai Kahl (<u>kahl.kai@mh-hannover.de</u>)
Tel.: +49-511-532-2495 / Fax.: +49-511-532-2415

Dr. Ivo Heitlandt (heitland.ivo-aleksander@mh-hannover.de)

Tel.: +49-511-532-7367/ Fax.: +49-511-532-7375)

#### Universität zu Lübeck

Klinik für Psychiatrie und Psychotherapie

Universität zu Lübeck Ratzeburger Allee 160

23562 Lübeck

PD Dr. Philipp Klein (philipp.klein@uksh.de)

Tel.: +49-451-500-98871

Dr. med. Bartosz Zurowski (bartosz.zurowski@uksh.de)

Tel: +49-451-500-98831

#### Universitätsklinikum Marburg

Klinik für Psychiatrie und Psychotherapie

Rudolf-Bultmann-Straße 8

35039 Marburg

Prof. Dr. Tilo Kircher (tilo.kircher@staff.uni-marburg.de)

Tel.: +49-6421-58-65200 / Fax: +49-6421-58-65197 Dr. Ina Kluge (ina.kluge@staff.uni-marburg.de)

Tel.: +49-6421-58-6219

#### Klinikum der Universität München

Klinik für Psychiatrie und Psychotherapie

Nußbaumstr. 7 80336 München

Prof. Dr. Frank Padberg (<u>frank.padberg@med.uni-muenchen.de</u>)

Tel.: +49-89 4400-53358 / Fax: +49 89 4400-53930

Dr. Matthias Reinhard (matthias.reinhard@med.uni-muenchen.de)

Tel.: +49-89 4400-55512

### Universitätsklinikum Tübingen

Allgemeine Psychiatrie und Psychotherapie mit Poliklinik

Calwerstraße 14 72076 Tübingen

Prof. Dr. Andreas J. Fallgatter (andreas.fallgatter@med.uni-tuebingen.de)

Tel.: +49-7071-29-84858 / Fax: +49-7071-29-5379

Dr. Christian Frischholz (christian.frischholz@med.uni-tuebingen.de)

Tel.: +49-7071-29-86015

### 2.3. Financial support

The study is supported by the **German Research Foundation** within the Program **Clinical Trials**.

### 2.4. Signature and Consent statement

I have read this protocol and agree to conduct the study in accordance with the study protocol, the current version of the Declaration of Helsinki, ICH-GCP Guideline (International Conference on Harmonization - Good Clinical Practice) and applicable national laws and regulatory requirements. I also agree to handle all information concerning this study confidentially.

I will ensure that all personnel involved in the study under my direction will be informed about the contents of this study protocol and will receive all necessary instructions for performing the study according to the study protocol.

### **Principal Investigator (PI):**

Prof. Dr. Eva-Lotta Brakemeier

| | Bratomie |
|------|-----------|
| Date | Signature |

I have read this protocol and agree to conduct the study in accordance with the study protocol, the current version of the Declaration of Helsinki, ICH-GCP Guideline (International Conference on Harmonization - Good Clinical Practice) and, applicable national laws and regulatory requirements. I also agree to handle all information concerning this study confidentially.

I will ensure that all personnel involved in the study under my direction will be informed about the contents of this study protocol and will receive all necessary instructions for performing the study according to the study protocol.

### <u>Charité – Universitätsmedizin Berlin</u>

| Prof. Dr. Philip | op Sterzer | |
|------------------|------------|-----------|
| 22.3 | .2021 | Alfhur |
| Date | <u> </u> | Signature |
| Prof. Dr. Stepl | han Köhler | |
| Date | <u> </u> | Signature |

I have read this protocol and agree to conduct the study in accordance with the study protocol, the current version of the Declaration of Helsinki, ICH-GCP Guideline (International Conference on Harmonization - Good Clinical Practice) and, applicable national laws and regulatory requirements. I also agree to handle all information concerning this study confidentially.

I will ensure that all personnel involved in the study under my direction will be informed about the contents of this study protocol and will receive all necessary instructions for performing the study according to the study protocol.

| Prof. Dr. Kai Kahl | |
|--------------------|-----------|
| Date | Signature |
| Dr. Ivo Heitlandt | |

Signature

**Medizinische Hochschule Hannover** 

Date

I have read this protocol and agree to conduct the study in accordance with the study protocol, the current version of the Declaration of Helsinki, ICH-GCP Guideline (International Conference on Harmonization - Good Clinical Practice) and, applicable national laws and regulatory requirements. I also agree to handle all information concerning this study confidentially.

I will ensure that all personnel involved in the study under my direction will be informed about the contents of this study protocol and will receive all necessary instructions for performing the study according to the study protocol.

### **Universität zu Lübeck**

| PD Dr. Philipp Klein | |
|----------------------|-----------|
| | Veen |
| Date | Signature |
| Dr. Bartosz Zurowski | |
| Date | Signature |

I have read this protocol and agree to conduct the study in accordance with the study protocol, the current version of the Declaration of Helsinki, ICH-GCP Guideline (International Conference on Harmonization – Good Clinical Practice) and, applicable national laws and regulatory requirements. I also agree to handle all information concerning this study confidentially.

I will ensure that all personnel involved in the study under my direction will be informed about the contents of this study protocol and will receive all necessary instructions for performing the study according to the study protocol.

| Universitätsklinikum Marburg | |
|------------------------------|---------------|
| Prof. Dr. Tilo Kircher | |
| <br>Date | <br>Signature |
| Dr. Ina Kluge | |

Signature

Date

I have read this protocol and agree to conduct the study in accordance with the study protocol, the current version of the Declaration of Helsinki, ICH-GCP Guideline (International Conference on Harmonization – Good Clinical Practice) and, applicable national laws and regulatory requirements. I also agree to handle all information concerning this study confidentially.

I will ensure that all personnel involved in the study under my direction will be informed about the contents of this study protocol and will receive all necessary instructions for performing the study according to the study protocol.

### Klinikum der Universität München

| Prof. Dr. Frank Padberg | |
|-------------------------|-----------|
| 22.03.2021 | FRE |
| Date | Signature |
| Dr. Matthias Reinhard | |
| Date | Signature |

I have read this protocol and agree to conduct the study in accordance with the study protocol, the current version of the Declaration of Helsinki, ICH-GCP Guideline (International Conference on Harmonization — Good Clinical Practice) and, applicable national laws and regulatory requirements. I also agree to handle all information concerning this study confidentially.

I will ensure that all personnel involved in the study under my direction will be informed about the contents of this study protocol and will receive all necessary instructions for performing the study according to the study protocol.

### **Universitätsklinikum Tübingen**

| Prof. Dr. Andreas J. Fallgatter | |
|---------------------------------|-----------|
| 22.03.2021 | Fallgatt |
| Date | Signature |
| Dr. Christian Frischholz | |
| Date | Signature |

# 3. Scientific Background

Up to one third of depressed patients develop persistent depressive disorder (PDD) with an estimated lifetime prevalence between 3% and 6% (Angst et al., 2009; Murphy & Byrne, 2012). Given the high degree of suicidality, comorbidity, and non-response to outpatient treatments (Murphy & Byrne, 2012; Bschor et al., 2014; Murphy et al., 2017; Köhler et al., 2019), many PDD patients require hospitalization as guidelines recommend; accordingly, about half of all psychiatric inpatients with depression suffer from PDD (Härter et al., 2004; Hölzel et al., 2010; Bschor et al., 2014; DGPPN et al., 2015; Köhler et al., 2016). In Germany, about 70.000 PDD patients are currently treated as inpatients per year, causing an enormous economic burden of an estimated 1 billion € annually. Thus, they constitute one of the main cost drivers for depression care (Luppa et al., 2007). However, for these inpatients no evidence-based treatment exists (Köhler et al., 2016; Schefft et al., 2019). Despite an overall reduction in depression with long psychotherapeutic inpatient treatment (Keller et al., 2001), PDD inpatients reach lower response rates, report higher treatment dissatisfaction, and are more likely to relapse after discharge than acutely depressed inpatients (Härter et al., 2004; Keller et al., 2001). Since most inpatients are non-responders to standard treatments, new treatment-phase programs combining acute and continuation treatments are urgently needed to overcome treatment-resistance (TR) (Köhler et al., 2016; Schefft et al., 2019). CBASP is the only psychotherapy specifically tailored for PDD (McCullough et al., 2014) demonstrating efficacy as outpatient treatment through a growing number of RCTs (Keller et al., 2000; Schramm et al., 2011; Wiersma et al., 2014; Michalak et al., 2015; Schramm et al., 2017; see Jobst et al., 2016 and Negt et al., 2016 for a review and meta-analysis). Thus, we modified CBASP as a manualized multimodal inpatient program for the severely ill PDD inpatients with TR (Brakemeier & Normann, 2012; Brakemeier, Guhn & Normann, in press). Our pilot studies indicate very good feasibility and promising outcome (Brakemeier et al., 2011; Brakemeier et al., 2015; Sabaß et al., 2018; Guhn et al., 2019). Therefore, a randomized controlled trial is now mandatory for testing the superiority of the inpatient CBASP program vs. an evidence-based psychotherapy such as cognitive behavioral therapy (CBT), the 'gold standard' in depression treatment. We chose a specific version of CBT – behavioral activation (BA) (Kanter et al., 2009; Martell et al., 2015) – since BA is at least as effective as standard CBT in severely depressed patients (Cuijpers et al., 2007; Dimidjian et al., 2006; Spates et al., 2006; Shinohara et al., 2013; Richards et al., 2016) while being easier to train and to implement in inpatient settings (Snarski et al., 2011). In addition, we will address the important psychotherapy research question: what works for whom and why? (e.g., Norcross & Wampold, 2011).

Moderator analyses will examine whether childhood maltreatment (Bernstein & Fink, 1998; Nemeroff et al., 2003; Brakemeier et al., 2018) and methylation of exon IV of the BDNF gene (Frieling & Tadić, 2013; Tadić et al., 2014) have an impact on the differential efficacy of the treatments. DNA methylation of the BDNF exon IV promoter region as an epigenetic mechanism will be assessed at baseline to address the dynamic changes of depressive symptoms and their treatment response. Epigenetic mechanisms are modulated by environmental stimuli and are adaptive to different disease stages (Menke und Binder, 2014). First evidence for epigenetic markers like BDNF as outcome predictor (in a pharmacotherapy depression trial) has been gathered (e.g., Frieling & Tadic, 2013; Lieb & Frieling, 2018). DNA methylation of one specific CpG located in the promoter region of BDNF exon IV has repeatedly been shown to accurately predict non-response to monoaminergic antidepressant drugs. As BDNF has been implicated in neurobiological processes fundamental to successful psychotherapy (ie. learning, memory, neural plasticity) it is reasonable to believe that

epigenetic (dys-)regulation of the BDNF gene might also play a role in response to psychotherapy and might therefore be useful as a prognostic marker. Apart from the BDNF system, (dys-)regulation of several genes have been proposed to be involved in neurobiological pathways underlying psychotherapeutic processes (e.g. Vinkers et al., 2021). Epigenome wide association studies as well as candidate gene studies are possible to detect new genetic loci involved (Vinkers et al., 2021). Machine learning algorithms integrating epigenome wide methylation data have been shown to be potent predictive tools for e.g. age acceleration ("epigenetic clocks") (e.g. Chaix et al., 2017)— in a similar way, it is likely that algorithms can be trained to learn based on the epigenome which therapy will suit best the individual patient's needs. Thus, in our study, blood samples for epigenetic analyses will be drawn to assess potential biomarkers for CBASP/BA response.

Regarding mediator analyses, we will investigate whether symptom improvements can be explained by an amelioration of interpersonal problems in CBASP (Horowitz et al., 2000; Jacobs & Scholl, 2005; Constantino et al., 2008; Klein et al., 2016) and an increase of activity levels in BA (Kanter et al., 2007; Rosenbaum et al., 2015; Forbes, 2020). A follow-up survey 48 weeks after the end of interventions will provide valuable results regarding the long-term success of the treatments.

Thus, the novel aspects of this trial are 1) comparing the multimodal CBASP inpatient program with a strong active comparator within treatment-resistant PDD patients by 2) applying a treatment-phase program while investigating 3) moderators and 4) mediators of change to guide personalized treatment and enable therapists to more specifically address psychotherapeutic needs of individual PDD patients in the future. Notably, 5) a costeffectiveness perspective further addresses health-economic issues and will enhance the relevance and potential benefit of CBASP (and BA) for public health (Drummond, 2007). Therefore, this trial will provide valuable information concerning allocation of resources (inpatient, dayclinic, and outpatient treatment) and may be of interest to decision makers in healthcare policy. Many hospitals in German-speaking (like Switzerland and Austria) and other countries (like USA, Denmark and Canada) already have implemented CBASP concepts. Due to the relatively short interventions, dose, and duration of the treatment-phase program, it is comparable to clinical practice, being at the same time affordable (for example by the German Health Care System). Notably, even in other countries the short inpatient intervention followed by dayclinic and outpatient treatment could be implemented. However, additional evidence needs to be provided before the CBASP inpatient program for treatment-resistant PDD is established on a broader scale influencing clinical practice. Thus, the results of this study have the potential to relieve the burden of this very serious and cost-intensive disease while improving human health.

# 4. Rationale and Hypothesis

### 4.1. Rationale

About half of all psychiatric inpatients with depression suffer from persistent depressive disorder (PDD). Given their high degree of treatment-resistance, comorbidity, suicidality, and hospitalization rates, this patient group appears to be particularly difficult to treat and, from a health economic perspective, constitutes a major challenge. The Cognitive Behavioral Analysis System of Psychotherapy (CBASP) is the only psychotherapy specifically tailored for PDD. Originally developed as an outpatient treatment, we have modified CBASP for the severely ill PDD patients with TR as a multimodal inpatient concept. Our pilot studies indicate

very good feasibility and promising outcome. Therefore, a randomized controlled trial is now mandatory for testing the superiority of the inpatient CBASP program vs. the evidence-based Cognitive Behavioral Therapy (CBT), the 'gold standard' in depression treatment. Behavioral Activation (BA) was chosen as the control intervention because BA, as a specific variant of CBT, is at least as effective as standard CBT in severely depressed patients while being easier to train and implement in inpatient settings. Both therapies will be applied as a treatment-phase program (10-week inpatient/ dayclinic acute treatment followed by 6-week outpatient continuation group-treatment) in combination with standardized and guideline-based pharmacotherapy. The proposed prospective, multi-center, randomized study with 396 PDD patients with TR will therefore address the primary research question: Is the CBASP program more effective than the BA program in this patient group? Our hypothesis is that after 16 weeks of treatment, CBASP will show a significant superiority over BA in reducing depressive symptoms. In addition, we will address the important psychotherapy research question: what works for whom and why? Moderator analyses will examine whether childhood maltreatment and methylation of exon IV of the BDNF gene have an impact on the differential efficacy of the treatments. Regarding mediator analyses, we will examine whether symptom improvements can be explained by an amelioration of interpersonal problems in CBASP and an increase of activity levels in BA. A follow-up survey 48 weeks after the end of the interventions will provide valuable results regarding the long-term outcome of the treatments.

Finally, the health economic potential of the interventions will be investigated through costbenefit analyses in order to provide important information on the cost-effectiveness of implementation in routine care for health policy. Thus, the results of this study will have the potential to relieve the burden of this very serious and cost-intensive disorder while improving human health. In addition, moderator and mediator analyses may guide personalized treatment and enable therapists to more specifically address psychotherapeutic needs of individual PDD patients in the future.

### 4.2. Hypothesis

It is hypothesized that CBASP (being tailored for the burdened subgroup of TR PDD inpatients) is significantly more effective than BA (being tailored for depression in general) after 16 weeks of treatment-phase programs (overall 20 individual and 26 group therapy sessions).

### 5. Study Design

This prospective, multi-center, randomized study with 396 TR PDD patients will compare the two manual-based inpatient programs CBASP (Brakemeier & Normann, 2012; Brakemeier, Guhn & Normann, in press) (as experimental intervention) and BA (Martell et al., 2015) (as control intervention).

To control group effects, we provide the treatment teams with precise study manuals for the CBASP- and BA-programs that describe all study treatments in detail. Since the risk of systematic errors is higher in inpatient psychotherapy studies than in outpatient studies due to more uncontrollable factors, we have done everything possible to minimize these uncontrollable factors, mainly by parallelization. Thus, the study manuals guarantee that both groups receive the same type, dose, and duration of study treatments, the same additional treatments, the same algorithm concerning medication, and the same dose of team training and supervision, etc. (see chapter 9). In addition, the study manuals clearly specify which

additional treatments are allowed for study patients. Furthermore, important conditions immanent in the inpatient setting also minimize confounding variables (such as same location and environment, same weather, same diet, same daily routine, same general hospital rules, same hospital climate, same chief physician, no or sparse interaction with family and friends, no work practice). In order to enable comparability of the participating sites and reduce a site effect, or a possible allegiance bias discriminating BA, the two interventions are carried out in each participating site on two separate specialized wards.

The sufficient sample size (N=396) and the six recruitment sites in different regions of Germany will assure generalizability of results and representativeness of the sample. Furthermore, we kept exclusion criteria to a minimum (expecting a high rate of comorbidity) to even enhance generalizability of our findings. Inclusion/exclusion criteria are specified to yield a population of PDD patients with a high degree of TR (see 8.2 and 8.3).

Power calculation for the proposed sample size of N=396 is based on a simulation study as recommended for linear-mixed effects models (Gelman & Hill, 2007). Please note that this estimate already takes into account that we expect about 14% missing data at the primary endpoint (i.e., after 16 weeks), because the simulation study already included assumptions about missing data. Concerning expected dropout rates, based on the RCT trial by Schramm et al. (2017), where 3% of patients dropped out immediately after randomization, we expect that about 5% of patients to drop out of the study immediately after randomization (no treatment and follow-up), although all efforts will be made during the informed consent procedure to include only patients who are willing to accept both arms and to continue study visits until W64/T5 (even if they drop out of treatment). In addition, in our one-arm pilot study (Brakemeier et al., 2015), 92.9% of the patients (65 out of 70) were fully compliant with the CBASP inpatient regime. Since in BA the same dose and duration of psychotherapy is scheduled we expect about 90% compliance in the multicenter trial in both groups. Therefore, we expect 95% x 90% = 85.5% of randomized patients to have HDRS-24 non-missing in week 16. Moreover, in our CBASP pilot study (Brakemeier et al., 2015), we observed only 12.9% losses to 6-months follow-up and 14.3% to 12 months follow-up. Therefore, we expect 15% of those who start treatment to have HDRS-24 missing in week 64, leaving 95% x 85% = 80.8% of those randomized with non-missing HDRS-24 in week 64.

We anticipate that about 1.000 patients have to be screened in order to randomize 396 patients (40% informed consent). In comparable studies slightly higher rates are found: in our own inpatient RCT study with depressed patients having received Electroconvulsive Therapy (ECT; Brakemeier et al., 2014) 61% informed consent and the RCT of Keller et al. (2000) 85% informed consent. The reason for why we are more conservative is that in the Brakemeier et al. (2014) trial the depressive patients while having been randomized had already successfully responded to inpatient treatment and were randomized to maintenance therapy. In the Keller et al. (2000) study all treatments were outpatient. PDD patients with TR who report for inpatient admission may be more difficult to motivate to participate in this inpatient RCT due to the severity and chronicity of the disease.

Regarding internal validity, group effects, the comparability of the sites, a site effect, or a possible allegiance bias discriminating BA, we have taken many precautions, as described in the following. Randomization with stratification for severity of depression (HDRS-24; Hamilton, 1960) and study site will be performed with an allocation ratio of 1:1. Due to the nature of interventions, blinding of patients/therapists concerning the treatment program is impossible, but all assessments as well as data analysis will be blinded to treatment allocation. Notably, patients are blinded to the study hypothesis by the Informed Consent process, as patients are told in the patient information and educational discussions about the study that

they will in any case receive one of two different scientifically based psychotherapy programs, although it is unclear which of the two programs is more effective; one program focuses on coping with interpersonal problems, the other on building up activities that seem important for personal life (see Informed Consent Form). Similarly, the members of the treatment teams of each study ward are not informed about the study hypothesis; however, they are informed that it has not yet been scientifically clarified which therapy is more effective.

Measures to ensure blinding will include locating the raters separately from the study wards, instructing patients not to mention information that could reveal their allocation, and providing back-up raters in case of unintentional unblinding. All blinded raters (student assistants at each participating site) will be trained in all instruments (HDRS-24, GAF, MINI-ICF, IMI-R, cost interview). Concerning HDRS-24, raters will be certified by a central rating of three videotaped HDRS-24 interviews. Additionally, the adherence and competence of the psychotherapists with regard to the specific CBASP or BA techniques will be evaluated regularly (measured with the observer-rated video-based CAR instruments). Since the patients will evaluate their subjective acceptance, satisfaction with and effectiveness of received treatments and the atmosphere of the ward etc. with the standardized questionnaire RevieW every week of treatment, we will also consider these subjective evaluations in our analyses (see 6.2).

## **Study Flow Chart**

Figure 2: Study Flow Chart



#### 6. Outcome Measures

### **6.1.** Primary Endpoint

The primary endpoint will be

 the change in HDRS-24 item score (Hamilton, 1960; Williams, 1988) from baseline to 16 weeks after randomization

The HDRS is considered being the "gold standard" as the most frequently used and well-validated clinician rated measure of depression severity (Carrozzino et al., 2020). As recommended by Carrozzino et al. (2020) we will use a semi-structured version of the 24 item version, including item definitions, anchor points and semi-structured interview questions. Each item is evaluated on a 3 to 5 level scale, for each of which a short description is given. The time frame of the asked symptomatology applies to the last week before the interview. On average, the processing time is 15 minutes. The range of the HDRS-24 is from 0 to 75. It is not recommended to make a diagnosis of depression based on cut-off value because the HDRS is primarily designed to be sensitive to changes and is therefore more suitable for measuring changes in the course. Most of the relevant trials we refer to use HDRS-24 change as primary outcome. The endpoint was set at week 16 after randomization, as CBASP is expected to show superiority over BA with a long duration and high dosage (see Cuijpers et al., 2010; Wiersma et al., 2014; Brakemeier et al., 2015; Schramm et al., 2017). HDRS-24 will be administered at screening (T0), week 1 (T1), 5 (T2), 10 (T3), 16 (T4), 64 (T5) by blinded observers being not otherwise involved.

### **6.2.** Secondary Endpoints, Moderators and Mediators

Secondary endpoints will be the following questionnaires and interviews:

- HDRS-24 (see above), assessed every second week and at week 64
- IDS-SR (Rush et al., 2000), assessed every second week and every second month during follow-up
- Brief Symptom Inventory (BSI; Derogatis & Spencer, 1993), assessed at week pre, 1, 5, 10, 16, and
- Global Assessment of Functioning (GAF; Hall, 1995), assessed at week pre, 1, 5, 10, 16, and 64
- World Health Organization Quality of Life (WHOQoL; Angermeyer et al., 2000), assessed at week pre, 1, 5, 10, 16, and 64
- Response (50% decrease on HDRS-24 score in comparison to baseline), remission (HDRS-24 of 10 or less on the HDRS-24), relapse rates (defined as rehospitalization for symptomatic worsening and/or a combination of an increase in HAMD 24 from discharge of equal or greater than 10 points and a current HAMD 24 score of equal or greater than 18 points), and dropout, assessed at week 5, 10, 16, and 64 (relapse-rate only at week 16 and 64)
- Cost interview (Wagner et al., 2014) assessed at week pre, 16, and 64; through the cost interview, the direct medical costs (inpatient stays, doctor's visits, emergency treatment, etc.), the direct non-medical costs (informal help, delinquent behavior, etc. and the indirect costs (days of incapacity to work, disability, unemployment) are recorded. In addition, a distinction is made as to whether the costs are due to mental disorders versus physical illnesses.

In addition, the following other important psychological variables will be assessed as further endpoints at week pre, 1, 5, 10, 16, and 64:

- Beck's Depression Inventory (BDI-II; Hautzinger et al., 2006)
- Brief Resilience Scale (BRS; Smith et al., 2008)
- Dysfunctional Attitude Scale (DAS; Hautzinger et al., 2005)

- Euthymia Scale (ES; Carrozzino et al., 2019)
- Experience in Close Relationships Scale Revised 8-item version (ECR-RD8; Ehrenthal et al., submitted)
- General Self-Efficacy Scale (GSE; Schwarzer & Jerusalem, 1995)
- Impact Message Inventory revised (IMI-R; Casper et al., 2000)
- Lübecker Questionnaire of Preoperational Thinking (LQPT; Kuehnen et al., 2011)
- Measure of disorders of capacity as defined by the International Classification of Function (Mini-ICF; Linden & Baron, 2005)
- Mental Pain Questionnaire (MPQ; Fava et al., 2019)
- Personality Inventory for DSM-5 Brief Form Plus Modified (PID5BF+ M; Kerber et al., submitted;
   Bach et al., in press)
- Rejection Sensitivity Questionnaire (RSQ; Downey & Feldman, 1996; Staebler et al., 2011)
- Revised-Green Paranoid Thoughts Scale (R-GPTS; Freeman et al., 2019)
- Social Network Index (SNI; Cohen, 1997)
- UCLA Loneliness Scale (UCLA; Döring et al., 1993; Russell, 1996)
- Well-being Index (WHO-5; Krieger et al., 2014)

The main moderators (measured at baseline) are:

- Childhood maltreatment measured by Childhood Trauma Questionnaire (CTQ; Bernstein et al., 2003; Wingenfeld et al., 2010)
- Epigenetic (Brain-derived neurotrophic factor (BDNF) methylation)

The main mediators (measured at baseline and week 1, 2, 4, 6, 8, 10, 12, 14, 16 and 64) are:

- Interpersonal problems (Inventory of Interpersonal Problems-revised, IIP-32-R, 32-item version;
   Horowitz et al., 2000)
- Activities (Behavioral Activation Depression Scale, BADS; actimeter-measured step-counts)

Finally, the following instruments are also applied to measure other important constructs

- Therapeutic relationship (Working Alliance Inventory, WAI; Wilmers et al., 2008) measured at week 1, 2, 4, 6, 8, 10, 12, 14, and 16)
- Subjective evaluation of important specific and unspecific working mechanisms of treatment (Review of last Week, RevieW; Koy, 2019; measured every week during the 16 weeks of treatment)

Nearly all measures have validated and are widely used, including the important CBASP or CBT/BA trials.

### 6.3. Further Endpoints

Safety will be assessed by monitoring adverse events, side effects and medication. (Severe) Adverse events (SAEs) and medication will be continuously monitored via a standardized questionnaire; negative effects including side effects of psychotherapy will be measured at

wk. 5, 10, 16, and 64 with the SEPIPS (Side Effects of Psychological Interventions Process Scale; Herzog et al., in prep.).

### 7. Methods of Data collection

The investigators are responsible for the performance of the trial in accordance with GCP guidelines and the study protocol as well as the correct data entry to the corresponding electronic case report form (eCRF). The self-reported questionnaires are completed by the patient herself/himself using tablets or computers electronically from the clinic and are thus directly integrated into the eCRFs. The study staff also enters the results of the clinical interviews directly into the eCRFs. The blood sample (approximately 10 ml) will be taken at the first study visit. Blood samples will be stored at the study centers and then transported twice a year to the central sample storage in the Hannover Unified Biobank (HUB). The blood will be evaluated in a study laboratory (Molecular Neuroscience laboratory at Hannover Medical School) regarding methylation of exon IV of the BDNF gene. The results are then entered into the eCRF by study staff. Blood respectively DNA samples will be stored for further exploratory genomic and epigenomic studies examining BDNF as a moderator for the response of depressed patients to methods of psychotherapy.

All patients will receive an actimeter to measure the number of steps during the entire study.

The data of the patients are documented with the EDC (Electronic Data Capture). The self-report questionnaires are entered directly by the patients. It should be noted that patients are invited to the clinic for all study visits so that they always use the certified equipment and study staff are always available to help with any questions. This will also contribute to a maximum good data quality. The data is entered directly into the eCRF via the web browser. As the system is a web application, a stable internet connection and an input device is required. Standardized input devices will be available to patients. Detailed instructions on how to use the EDC system are listed in the EDC manual, which is part of the ISF.

Furthermore, all individual psychotherapeutic sessions will be videotaped (including sound) by standard video cameras for 1) supervision purposes, 2) conducting the CAR ratings (assessment of adherence and competence) and 3) research purposes in the field of psychotherapy process research. Standardized evaluation methods are used to assess which processes take place in the therapy sessions and how these processes are related to the therapy outcome.

### Selection of patients

The investigators will keep a record of all study candidates who were considered for enrollment including screening failures that were never enrolled. A screening log form will be filed in the ISF.

## 8. Study Population

### **8.1.** Treatment groups

The study population consists of psychiatric inpatients with persistent depressive disorder who have been treatment-resistant. In total, the sufficiently large sample size (N=396) recruited at six participating sites in different regions of Germany (with a shared amount of patients) will assure generalizability and representativeness of results. Furthermore, we kept exclusion criteria to a minimum (expecting a high rate of comorbidity) to even enhance

generalizability of our findings. Inclusion/exclusion criteria are specified to yield a population of PDD patients with a high degree of TR.

#### **Patient recruitment**

The screening of the patients will be performed in the participating study sites. The recruitment of patients is supported by advertising measures, which will be produced between August and October 2020. For example, flyers will be sent and distributed to therapists in outpatient and inpatient practice and a website set up especially for the study will provide information about the study. Advertisements for the study will also be placed on other relevant websites (e.g. 'Deutsche Depressionshilfe', CBASP Network, etc.). It is expected that screening of 1.000 persons will result in 396 patients eligible for the study. The recruitment period will last for 30 months.

### 8.2. Inclusion criteria

- Age range: 20-70 years
- Primary DSM-5 diagnosis of PDD (300.4, 296.2x, 296.3x)
- Total HDRS score (24-item version) ≥ 20 at screening visit
- TR: Treatment-resistance defined as a level of 3 or higher on the Antidepressant Treatment
   History Form Short-Form (ATHF-SF; Sackeim et al., 2019) or medication intolerance or one
   psychotherapy (at least 25 sessions in the current episode conducted by a certified therapist)
- Sufficient knowledge of the German language
- Written informed consent

#### 8.3. Exclusion criteria

- Bipolar I or II disorder, active substance use disorders (abstinence shorter than 6 months), schizophrenia spectrum and other psychotic disorders, or antisocial personality disorder (all according to DSM-5)
- Acute suicidality
- Previous CBASP or BA treatment within the last year
- Inability to tolerate CBASP or BA (e.g., organic brain disorders, severe cognitive deficits)
- Inability to participate in dayclinic or continuation treatment

### 8.4. Methods against bias

#### 8.4.1. Randomization

Randomization with stratification for severity of depression and participating site with an allocation ratio of 1:1 will be performed by a blinded statistician. To ensure allocation concealment, only the leading investigator at each site will see the result of the allocation. This procedure is intended to minimize the bias due to allocation concealment. The

randomization of an eligible patient can only take place if **all** inclusion criteria and **none** of the exclusion criteria are fulfilled.

The group assignment is based on random permuted blocks with random block sizes and stratification for severity of depression (binary) and participating site. Regarding the severity of depression, an HRSD-24 score of at least 27 points was chosen as the binary cut-off criterion, since in the study by Schramm et al. (2017) the mean value of the HRSD-24 scale at the beginning of the study was also 27 points. Stratified permuted blocks ensure balance between both treatment groups, the balance within each participating site, and balance of the major covariate (depression severity). The use of random block sizes ensures that the next randomization assignment cannot be guessed.

#### 8.4.2. Blinding

Due to the nature of interventions, blinding of patients/therapists concerning the treatment is impossible. However, the patients/treatment team on the wards will be blinded regarding the primary study hypothesis (see 4.2) because the patients and the treatment teams will be told that it is not yet known which of the two psychotherapy programs is more effective in treating PDD patients with TR. In addition, the clinical raters (thus, all assessments) and the trial statistician (thus, the data analysis) will be blinded to treatment allocation during the analysis of the primary outcome. Ideally, the same clinical rater (student assistants at each participating site) will rate the patient at all measurement times. Procedures to ensure blinding will include locating the clinical raters separately from the study wards, instructing patients not to mention information that could reveal their allocation, and providing backup raters in case of unintentional unblinding. All blinded clinical raters will be trained in all instruments (HDRS-24, GAF, MINI-ICF, IMI-R, cost interview). Concerning HDRS-24, the raters are first trained through a three-hour (web-based) training session and then complete an evaluation of three standardized videotaped HDRS-24 interviews. Only if they have successfully completed these three ratings (which means that the difference is less than 3 points for each rating), they will be admitted as study raters. Strict concealment of randomization will be guaranteed to exclude selection bias (see 8.4.1). Since randomization of therapists is impossible, demographic and professional characteristics of therapists will be assessed (instrument: THAT; Klug et al., 2002).

### 8.4.3. Control of therapy allegiance

Therapy allegiance, i.e. treatment preference of the investigators or therapists, has been discussed as an important influencing factor for results in psychotherapy research (Luborsky et al., 1999; Munder et al., 2013; Robinson, Berman & Neimeyer, 1990). Thus, several procedures have been implemented to minimize the allegiance effect:

- 1. Several investigators have been involved in the design of this study who represent a "mix of therapy allegiances".
- 2. The two interventions are carried out in all sites with the same lengths and duration.
- 3. The entire treatment team of each study ward will be trained and supervised either in BA or in CBASP by highly experienced CBASP/BA experts. Before study start, all 12 wards of the six participating sites will be trained (intensive training workshops, same amount for both arms) in one of the two concepts and fresh-up team trainings for both arms will be performed every six months. The same amount of training and supervision for each study ward will be offered

with the possibility that rather unexperienced BA wards receive more training/supervision inter alia by our BA experts. In addition, training on-site visits of the core team of less experienced sites on an experienced BA ward will be organized.

#### **8.4.4.** Control of overlapping treatments

The following measures will be taken to prevent confounding of treatment conditions through the overlap of treatment methods:

- All study therapists are obligated to adhere to the therapeutic procedures and interventions described within the manuals. In addition, treatment fidelity, adherence and competence will be assessed: Trained study assistants will rate videotapes of 1 individual therapy session of each study patient on a random basis under supervision of the trial site psychologists. s. In addition, a separate team of the experts will randomly evaluate one videotaped individual session of each patient. Before treating study patients, the psychotherapists have to meet the criteria for mastery of CBASP or BA procedures as assessed by evaluation of their performance. The competence and adherence observer ratings for both individual and group sessions are oriented towards the already established assessment for cognitive therapy - the Cognitive Therapy Scale (CTS; Weck et al., 2010) - and are based on adherence scales for CBASP and BA that have already been used in other studies. We call our adapted instruments CBASP-CAR (Observer-based Competence and Adherence Rating of CBASP) and BA-CAR (Observer-based Competence and Adherence Rating of BA). The CAR evaluations refer to the therapeutic approach and the respective strategies of the two treatments (CBASP, BA). Hence, we will determine a minimum cut-off that reflects the demands on adherence of therapists. All values above the minimum cut-off will record therapist's competence on the scale. In addition, after each session the therapist (both individual and group therapists) will fill out a check list regarding the employed interventions. The validity of the therapist statements will be checked through external assessment of the video recordings. In posthoc analysis it will be checked if the expected differences regarding intervention characteristics appear within the two therapies.
- The two interventions are carried out on two separate specialized wards. Each study therapist will be involved in only one of the two psychotherapy programs and will accordingly only perform one of the two psychotherapies.
- To evaluate therapist attitudes towards CBASP and BA, questionnaires will be applied at the therapy training, after the first study patient, and after study termination.
- Possible influences through qualification differences of the therapists will be controlled as follows
  - All therapists have completed professional training or are in their at least second training year (out of three) for certification as licensed psychotherapist.
  - All therapists have completed a comprehensive training (at least 24 UE) within the respective treatment approach. All therapists will conduct two pilot cases with at least 8 sessions supervised by at least 3 sessions.
  - Concerning their influence upon the efficacy of treatment, level of training and professional experience of the therapists will be collected and reviewed.

### **8.4.5.** Control of confounding factors

- The influence of the trial site upon efficacy of the respective treatment approaches will be investigated as a separate factor.
- Patients will be asked not to engage in off-study psychosocial or psychiatric interventions during the 16 weeks of treatment period.

#### 8.4.6. Control of measurement bias

- All clinical raters will have completed (web-based) training for rating HRSD.
- Guidelines for all rating scales are available.
- The interrater reliability will be determined on the basis of at least 3 recorded HRSD ratings.

## 9. Study Procedure

## 9.1. Study visit overview

The following Table 2 summarizes the proposed frequency and scope of trial visits including all instruments and the duration of post-trial follow-up, as well as the six main measurement time points (T), and 17 trial visits (V).

Table 2: Frequency and scope of trial visits

| | Screening | Inpatient I | | | Inpatient II/Dayclinic | | | Continuationphase | | | Naturalistic follow-up | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Main Measurement Timepoints (T) | T0 | T1 | | | T2 | | | T3 | | | T4 | | | | | | T5 |
| Trial Visits (V) | V1* | V2 | V3 | V4 | V5 | V6 | V7 | V8 | V9 | V10 | V11 | V12 | V13 | V14 | V15 | V16 | V17 |
| Week | pre | 1 | 2 | 4 | 5 | 6 | 8 | 10 | 12 | 14 | 16 | 24 | 32 | 40 | 48 | 56 | 64 |
| Informed Consent | х | | | | | | | | | | | | | | | | |
| Random** | х | | | | | | | | | | | | | | | | |
| In-/Exclusion criteria | х | | | | | | | | | | | | | | | | |
| Patients master data | х | | | | | | | | | | | | | | | | |
| Patient preference | х | | | | | | | | | | | | | | | | |
| ATHF / concomitant medication | x | | | | | | | | | | | | | | | | |
| DIPS | х | | | | | | | | | | x | | | | | | х |
| SCID-5-PD | х | | | | | | | | | | х | | | | | | х |
| Primary Efficacy | | | | | | | | | | | | | | | | | |
| HDRS-24*** | х | х | | | х | | | х | | | Х | | | | | | х |
| Key secondary endpoints | | | | | | | | | | | | | | | | | |
| HDRS-24*** | х | х | х | x | | х | х | х | х | х | x | | | | | | х |
| IDS-SR | х | х | х | х | | х | х | х | х | х | х | х | х | Х | х | х | х |
| BSI, GAF***, WHOQOL | х | х | | | х | | | х | | | х | | | | | | х |
| Response, remission, dropout-rate | | | | | х | | | х | | | х | | | | | | х |
| Relapse-rate | | | | | | | | | | | х | | | | | | х |
| Cost Interview | х | | | | | | | | | | х | | | | | | х |
| Further endpoints | | | | | | | | | | | | | | | | | |
| BDI-II, BRS, BSI, DAS, ECRRD8, ES, GSE,<br>IMI-R***, LQPT, MINI-ICF**, MPQ | x | x | | | x | | | x | | | x | | | | | | x |
| PID5BF+M, RSQ, R-GPTS, SNI, UCLA,<br>WHOQoL, WBI | | | | | | | | | | | | | | | | | |
| Moderators of Change | | | | | | | | | | | | | | | | | |
| CTQ, BDNF methylation | х | | | | | | | | | | | | | | | | |
| Mediators of Change | | | | | | | | | | | | | | | | | |
| IIP-32-R, BADS, Step counts | х | х | x | х | | x | x | x | х | x | x | | | | | | х |
| Side effects /( Serious) Adverse events | | | | | | | | | | | | | | | | | |
| SAEs and medication | | х | х | х | х | х | х | х | х | х | х | | | | | | х |
| SEPIPS | | | | | х | | | х | | | х | | | | | | х |
| Therapeutical Relationship, Adherence- and Competence Rating, Subjective Evaluation of Important Domains, Therapist | | | | | | | | | | | | | | | | | |
| WAI, CBASP-CAR***, BA-CAR*** | | х | х | х | х | х | х | х | х | х | х | | | | | | |
| RevieW**** | | х | х х | х | х | х х | х х | хх | хх | х х | хх | | | | | | |
| THAT | | х | | | | | | | | | | | | | | | |

**Note.** Primary endpoint is marked red; \* V1 is divided into V1a to V1d (see Figure 3); \*\* Randomization will be performed between T0/V1 and T1/V2; \*\*\* Blinded observer ratings; \*\*\*\* Two crosses per cell because the questionnaire RevieW is done weekly

#### 9.2. Visit 1

Visit 1 (T0) is divided into Visit 1a - 1d and takes place during the screening phase. A detailed plan is shown in Figure 3.

- Visit 1a can be carried out as a telephone or personal screening and lasts 20 30 minutes; the
  patient is informed about the study and the patient information is handed out or sent to
  her/him; inclusion and exclusion criteria are requested by a structured screening process
- Visits 1b, 1c and 1d should follow each other as soon as possible (maximum interval of 1 week)
- At the beginning of Visit 1b the patient should agree to participate in the study (informed consent).
- In Visits 1b and 1c the corresponding interviews are conducted by the blinded rater (see Fig. 3)
- Between the Visits 1b and 1c, patients are asked to fill in the questionnaires at home on a tablet or computer; this work can also be interrupted and resumed later or on a following day; if the patients do not have a computer or tablet, they can complete the questionnaires after or before the study visits using standardized input devices provided by the study site.
- If the patient has agreed to participate in the study (informed consent) in Visit 1b and has also been identified as suitable with regard to the inclusion and exclusion criteria, before visit 1d the randomization will be performed by a blinded statistician and this information is given to the patient at visit 1d; the date for admission on the ward will be fixed.

Figure 3: Detailed Screening Flow



#### 9.3. Visit 2-5

- Visits 2-5 take place during the inpatient phase I
  - Visits 2 within the first two days after admission (week 1)
  - Visits 3 and 4 at the end of weeks 2 and of the inpatient treatment
  - Visit 5 at the last or penultimate day of the inpatient phase
- Conduction of the corresponding instruments (see Table 2)
- Visit 2 and 5 are main measuring points (T1 and T2)

### 9.4. Visit 6-8

- Visits 6-8 take place during the inpatient phase II / dayclinic phase
  - Visits 6-7 at the end of weeks 6 and 8 of the inpatient phase II / dayclinic phase
  - Visit 8 at the last or penultimate day of the inpatient phase II / dayclinic phase
- Conduction of the corresponding instruments (see Table 2)
- Visit 8 is a main measuring point (T3)

#### 9.5. Visit 9-11

- Visits 9-11 take place during the continuation phase
  - Visits 9 and 10 at the end of weeks 12 and 14 of the continuation treatment
  - Visit 11 at the last or penultimate day of week 16 (last week of the continuation phase)
- Conduction of the corresponding instruments (see Table 2)
- Visit 16 is the main measuring point (T4, primary outcome)

### 9.6. Visit 12-17

- Visits 12-17 take place during the naturalistic follow-up.
  - Visits 12-16 at the end of weeks 24, 32, 40, 48, and 56 of the naturalistic follow-up
  - Visit 17 at the last or penultimate day of week 64 (last week of the naturalistic follow-up)
- Conduction of the corresponding instruments (see Table 2)
- Visit 17 is a main and the last measuring point (T5)

### 9.7. Conduction of the Interventional Arm (CBASP)

The CBASP program will follow a strict standardized treatment manual being based on (Brakemeier & Normann, 2012; Brakemeier, Guhn & Normann, in press).

During the 5-week inpatient phase I and the 5-week inpatient phase II / dayclinic treatment the patient will receive the following CBASP treatments per week:

- 2 individual therapy sessions (duration: 50 min per session)
- 2 group therapy sessions (duration: 100 min per session)

- 1 nurse contact (therapeutic exchange with a nurse) (duration: 25 min per contact)
- 1 exercise therapy (duration: 75 min per therapy)

During the 6-week outpatient treatment the patient will receive the following CBASP treatment per week:

1 group therapy session (duration: 100 min per session)

All individual sessions will be videotaped (including sound) for supervision purposes, for conducting the CAR ratings (assessment of adherence and competence) and for research purposes in the field of psychotherapy process research. Standardized evaluation methods are used to assess which processes take place in the therapy sessions and how these processes are related to the therapy outcome.

In addition, the following workshops and supervisions are conducted for the CBASP treatment team:

- one start-up site workshop before study start conducted for the entire treatment team by one of the following CBASP experts: Prof. Dr. E.L. Brakemeier, Dr. A. Guhn; PD Dr. J.P. Klein, Prof. Dr. S. Köhler; duration 9 hours (12 UEs)
- one start-up expert workshop before study start (after the start-up site training workshop) conducted for 4 participants per site (overall 24) by John Swan and Marianne Liebing-Wilson; duration 9 hours (12 UEs)
- fresh up training every six months conducted by one of the following CBASP experts: Prof. Dr. E.L.
   Brakemeier, Dr. A. Guhn; PD Dr. J.P. Klein, Prof. Dr. S. Köhler; duration 9 hours (12 UEs)
- weekly CBASP supervisions by a site supervisor for all individual therapists; duration 60 minutes
- every second month CBASP team supervisions by external experts (one of the following persons:
   Prof. Dr. E.L. Brakemeier, Dr. A. Guhn; PD Dr. J.P. Klein, Prof. Dr. S. Köhler); duration 120 minutes

#### 9.8. Conduction of the Control Arm (BA)

The BA program will follow a strict standardized treatment manual being based on (Martell et al., 2015).

During the 5-week inpatient phase I and the 5-week inpatient phase II / dayclinic treatment the patient will receive the following BA treatments per week:

- 2 individual therapy sessions (duration: 50 min per session)
- 2 group therapy sessions (duration: 100 min per session)
- 1 nurse contact (therapeutic exchange with a nurse) (duration: 30 min per contact)
- 1 exercise therapy (duration: 75 min per therapy)

During the 6-week outpatient treatment the patient will receive the following BA treatment per week:

1 group therapy session (duration: 100 min per session)

All individual sessions will be videotaped for supervision purposes, for conducting the CAR ratings (assessment of adherence and competence) and for research purposes.

In addition, the following workshops and supervisions are conducted for the BA treatment team:

- one start-up site workshop before study start conducted for the entire treatment team by one of the following BA experts: Dr. E. Fassbinder, Prof. Dr. K. Kahl, Prof. Dr. U. Schweiger; duration 9 hours (12 UEs)
- one start-up expert workshop before study start (after the start-up site training workshop)
   conducted for 4 participants per site (overall 24) by Prof. Dr. J. Kanter, duration 9 hours (12 UEs)
- fresh up training every six months conducted by one of the follwing BA experts: Dr. E. Fassbinder,
   Prof. Dr. K. Kahl, Prof. Dr. U. Schweiger; duration 9 hours (12 UEs)
- weekly BA supervisions by a site supervisor for all individual therapists; duration 60 minutes
- every second month BA team supervisions by external experts (one of the following persons: Dr. E. Fassbinder, Prof. Dr. K. Kahl, Prof. Dr. U. Schweiger); duration 120 minutes

### 9.9. Concomitant Therapy

To control group effects, it is clearly defined which additional treatments/services are permitted and which are prohibited for study patients (see Table 3). To control group effects, it is clearly defined which additional treatments/services are permitted and which are prohibited for study patients. With the permitted treatments/services, strict attention must be paid to ensuring that study patients in both treatment groups participate equally (parallelization).

**Table 3:** Permitted and prohibited treatments/services

| | Permitted (if performed in parallel for both study groups) | Prohibited |
|---|---|---|
| Inpatient<br>treatment<br>phase I<br>(5 weeks) | standardized physiotherapy group<br>(up to 3/week) | Mindfulness-based groups offered by therapists |
| | standardized occupational therapy group (up to 3/week) | All further psychotherapeutic or non-<br>psychotherapeutic group offers or individua<br>sessions |
| | algorithm-based study medication* | 3633.0.13 |
| | Crisis talk | |
| | Only if absolutely necessary for daily structure and performed in parallel for both study groups | |
| | relaxation-group | |
| | mindfulness-based offered by nurses | |
| | patient café | |
| | excursion | |
| | morning exercise | |

| | patient group | |
|---|---|---|
| | Permitted (if performed in parallel for both study groups) | Prohibited |
| | standardized physiotherapy group<br>(up to 3/week) | Mindfulness-based group offered by therapists |
| | standardized occupational therapy group (up to 3/week) | |
| | algorithm-based study medication* | |
| Inpatient<br>treatment<br>phase II or<br>dayclinic<br>treatment<br>(5 weeks) | Only if absolutely necessary for daily structure and performed in parallel for both study groups | All further psychotherapeutic or non- |
| | relaxation- or mindfulness-based group offered by nurses | psychotherapeutic group offers or individual sessions |
| | patient café | |
| | excursion | |
| | morning exercise | |
| | patient group | |
| | Permitted | Prohibited |
| Outpatient<br>treatment<br>6 weeks | algorithm-based study medication* | All further treatments by the clinic/ward |
| | If possible in these 6 weeks, outpatient psychotherapy should pause | |

### \*Medication add-on treatment

Most patients will be on medication at study entry due to the severity of illness. All patients will receive an optimized, algorithm-based antidepressant medication following the current S3-Guidelines on Unipolar Depression (DGPPN et al., 2015; Middleton et al., 2005). In case of nonresponse:

- 1st line dose escalation (if appropriate)
- 2nd line lithium augmentation
- 3rd line augmentation with 2nd generation antipsychotics or evidence-based combinations of antidepressants
- 4th line change of antidepressant.

Only the following psychopharmacological rescue medication may be prescribed during the course of the study:

 Zopiclone (on demand up to 7.5 mg/day orally) or Quetiapine (on demand up to a dose of 50 mg/day orally) for sleep disturbances.
Promethazine (on demand up to 75 mg/day orally) or Quetiapine (on demand up to 50 mg/day orally) for agitation.

After discharge from inpatient setting or dayclinic, all patients will continue on their last medication, which may be further optimized according to the S3-Guideline (DGPPN et al., 2015) if needed during continuation treatment. Medication is documented in the eCRFs and will be treated as covariates in the final efficacy analysis.

## 9.10. Study Sites

The participating sites that were selected by the Coordinating Investigator have adequate staff and experience in treating overall 400 patients and in conducting clinical studies with the same or similar indications. The participating sites include experienced psychotherapists and physicians and supportive staff with adequate time, the targeted patient population and technical expertise to complete the protocol.

# 9.11. Treatment after end of study

After the end of the study treatment (i.e. after 16 weeks) a naturalistic follow-up takes place for 48 further weeks (12 months). During this time, due to the naturalistic character patients may receive any therapy, but CBASP patients should not receive BA therapy and BA patients should not receive CBASP therapy. After the end of the study (i.e. after the follow-up), patients can receive the other treatment if they are interested and indicated, whereby study staff will help to arrange appropriate CBASP or BA treatment places (inpatient or outpatient).

# 9.12. Study Schedule

### Schedule

- Recruitment period (months): 30
- Study treatment per patient (days): 112 (16 weeks)
- Study duration per patient (days): 448 (64 weeks, incl. follow-up)
- First patient in to last patient out (months): 34 (without follow-up), 46 (incl. follow-up)
- Duration of the entire study (months): 58

End of the study is defined as "Last Patient Out" and database closure.

In the Figure 4 the preparation, pre-trial visits to and initiation of sites, recruitment, follow-up, data cleaning/analysis, and amount of funding required at each milestone is summarized.

**Figure 4:** Diagram reflecting the preparation, pre-trial visits to and initiation of sites, recruitment, follow-up, data cleaning/analysis, and amount of funding required at each milestone



## 10. Add-on Studies

In the following, two add-on studies are described, which are used to investigate further mediators and mechanisms of change of the two treatment programs. After consenting to the main ChangePDD study, the patients are informed about these two add-on studies and can then decide whether they want to participate in one or both of the additional studies. Participation in these add-on studies is therefore not obligatory for the study patients but optional. Thus, the two studies are described separately in this chapter 10. In order to get an overview of the design and the instruments when patients participate in both add-on studies in addition to ChangePDD, we have adapted Table 2 and Figure 3 accordingly (see 10.3).

## 10.1. ChangePDD-EMA

In this add-on study, in addition to the questionnaire-based measurement of symptoms described above (see chapter 6), data on affect, interpersonal behavior, social context, and loneliness are collected using an EMA (Ecological Momentary Assessment) approach. Responsible for this add-on study are Prof. Dr. Stephan Köhler, Dr. Anne Guhn, Prof. Dr. Johannes Zimmermann, Dr. Tim Kaiser, Prof. Dr. Philipp Sterzer and Prof. Dr. Eva-Lotta Brakemeier. As already mentioned, participation in this supplementary study is optional and does not influence inclusion in the main ChangePDD study. The add-ons to the regular study design and data analysis are described below.

### **10.1.1** Theoretical motivation

Compared to healthy controls and patients with episodic depression, PDD patients report more hostile-submissive interpersonal styles (Bird et al., 2018). However, there has been less research on the "in-the moment assessment" of social experiences in patients in PDD with regard to dynamic interplay of affect, interpersonal behavior and social context. Ecological Momentary Assessment (EMA) provides an ecologically valid tool to monitor daily experiences and its influence on social interaction. Recent research indicates a close relationship between

negative affective experiences during social interactions and the perceived effectiveness and enjoyment of those experiences at the end of the day (Geyer et al., 2018). In addition, a recent non-controlled CBASP study reports less loneliness after 10 weeks of inpatient CBASP (Reinhard et al., accepted). To what extent this is specific to CBASP or will also be a concomitant effect in BA warrants investigation.

The ChangePDD trial is particularly suitable to target the assessment of social interactions and behavioral activation in PDD patients as well as treatment change through therapeutic strategies that target both social interactions (CBASP) and mobility (BA). By the use of a smartphone application, participants are asked daily short questions about their current mood, interpersonal strength, behavioral activation/avoidance, social stress, and feelings of loneliness. This will be done over the course of the *ChangePDD* trial starting one week before admission to the ward and ending one week *after* the end of the outpatient treatment (see figure 5).

## 10.1.12 ChangePDD-EMA study design

In addition to data collection of the main mediators described above (see 6.2: IIP-32-R, BADS and actimeter-measured step count) collected during the treatment phase within ChangePDD (see Table 2), this add-on study will collect EMA data during three phases: 1) 1 week pretreatment, 2) 16 weeks of ChangePDD treatment, 3) one week post-treatment (total 18 weeks of EMA data collection). During the pre- and post-treatment weeks, 5 assessments per day are conducted and during the main study phase only one assessment per day is conducted (see Figure 5).

Figure 5: Study Design ChangePDD-EMA



Patients will be informed about this add-on study ChangePDD-EMA during study visit 1c, where they will sign the informed consent.

The assessment will be conducted via the app "Ethica". The app "Ethica" is DSGVO-compliant. The encryption matches a standard in the industry according to the producers. There will be a strict anonymization of the data with a clear division between personal data (meta data; accessible only by personnel for technical purposes) and study data (anonymous; accessible only by scientists). Participants are able to withdraw their consent at any point, resulting in the elimination of their data. At no point in time will assessed data be passed on to third parties. The servers on which the data is stored are located in Canada. A detailed description of the data protection concept can be found on the provider's website:

<u>https://ethicadata.com/legal#privacy-policy</u>. Several scientific EMA-studies have been conducted via this program worldwide and in Europe.

Furthermore, the app "Ethica" is compatible with Android and Apple and will be installed on the patients smartphone after their informed consent. After completing the study it will be deleted.

## 10.1.2 ChangePDD-EMA data assessment and analysis

The Interpersonal-Activation-Diary (IAD) was developed following Zimmermann et al. (2019) for this add-on study and consists of 23 items (see Table 4). These domains, which include interpersonal strength, behavioural activation/avoidance, social stress, and loneliness are hypothesized to be mechanisms of change especially of CBASP (interpersonal strength, social stress, loneliness) and of BA (behavioural activation/avoidance).

During the pre- and post-treatment weeks there will be 5 times daily request for data entry between 10 a.m. and 8 p.m.

- First to fourth survey
- a) 1 item on mood: How are you currently feeling? Response format: visual analogue scale with the poles very bad very good)
- b) 1 item on social context: Where are you right now? Response options: I am alone, I am with a family member, my partner, my colleagues, a friend or acquaintance)
- The last (5th) survey (8 p.m.): IAD + (+ = plus three items).

During the ChangePDD treatment phase the assessment will be once a day in the evening (e.g. 8 p.m.) containing the IAD.

**Table 4** Item overview of the Interpersonal-Activation- Diary (IAD)

| No. | Construct | Item* |
|---|---|---|
| | Interpersonal Strength | |
| 1 | "Connect" | I liked being with other people. |
| 2 | "Engage" | I was more outgoing, in order to get in touch with others. |
| 3 | "Lead" | I was able to ask other people for what I wanted. |
| 4 | "Direct" | I could fend for myself. |
| 5 | "Balance" | I was able to say "no" to others. |
| 6 | "Restrain" | I was able to listen and think before acting in relationships. |
| 7 | "Cooperate" | I was cooperative. |
| 8 | "Consider" | I felt enriched when I was able to help others. |
| | Activation-Avoidance | |
| 1 | Activation 1 | I was an active person and achieved the goals I set for myself. |

| 2 | Activation 2 | I made good decisions regarding which activities I partake in and which situations I seek out. |
|---|---|---|
| 3 | Activation 3 | I did many and different activities. |
| 4 | Activation 4 | am content with the kind and number of activities I did. |
| 5 | Activation 5 | lid things I enjoy. |
| 6 | Avoidance 1 | as mainly focused on avoiding uncomfortable things or fleeing from them. |
| 7 | Avoidance 2 | here were things to do, which I did not complete. |
| 8 | Avoidance 3 | spent a lot of my time thinking about my problems again and again. |
| | Social Stress | |
| 1 | Social Stress | I was ignored, dismissed or rejected by others. |
| 2 | Social Stress | I was let down by a person close to me. |
| 3 | Social Stress | I was accused, criticized or talked down by someone. |
| 4 | Social Stress | I was used or betrayed by someone. |
| | Loneliness | ess |
| 1 | Loneliness | I was alone or had little social contacts. |
| 2 | Loneliness | I felt lonely today. |
| 3 | Loneliness | I felt excluded today. |

<sup>\*</sup>Note: eight items each on interpersonal strength and behavioral activation and avoidance four items on social stress (modified according to Zimmermann et al., 2019) with the addition of another item on loneliness from the Personality Dynamics Diary (PDD; Zimmermann et al., 2019) as well as two items on loneliness from the Psychological Item Pool for Corona Outbreak (PIPCO; Buecker et al., 2020).

## **Data Analysis**

All data assessed in the context of the ChangePDD-EMA Add-on study will be analyzed using Dynamic Structural Equation Models (Asparouhov et al., 2018).

#### 10.2. Effort Task

In addition to the goals of the ChangePDD study, in this add-on study moderators and mediators of change of **BA** are examined. These mediators and moderators will be assessed by means of combining a behavioral effort task with computational modelling, allowing us to estimate mechanisms underlying depressive symptoms and processes assumed to lead to change due to BA. The task and design could also allow us to identify predictors of response to BA on an individual patient level. Dr. Isabel Berwian, Prof. Henrik Walter, Prof. Quentin Huys and Prof. Eva-Lotta Brakemeier are responsible for this add-on study. As already mentioned, participation in this supplementary study is optional and does not influence inclusion in the main ChangePDD study.

## 10.2.1 Theoretical motivation and hypotheses

Patients with depression show reduced engagement in rewarding activities (APA, 2013). The decision to engage in rewarding activities (e.g. going out, meeting friends) compared to "depressive" behaviors (staying in bed) can be viewed as a trade-off between the anticipated reward and the anticipated effort for each behaviour (Berwian et al., 2020). The reduction in rewarding activities seen in depression might hence result from decreased anticipated reward or from increased anticipated effort. Behavioral Activation (BA), a widely disseminated first-line therapy for depression (Lewinsohn, 1974; Nagy et al., 2020) contains component interventions that aim to directly address these aspects: planning, scheduling and monitoring of rewarding activities. The aim of planning is to ensure activities are realistic and achievable, thereby reducing the probability that effort will be spent without achieving a goal. The aim of scheduling rewarding activities is to ensure rewards are experienced. Finally, monitoring one's responses and feelings after rewarding activities helps to compare it to earlier expectation of effort and reward. The underlying assumption is that the experience of successful planning and rewarding activities re-establish reward and effort expectations.

These theoretical assumptions lead to the following two core hypotheses: 1) Experience of reward or effort moderates and predicts response to BA.

2) Anticipation of effort or reward is a mediator of this response.

As a secondary hypothesis, we suggest:

1) The above effects are stronger in patients receiving BA compared to patients receiving CBASP.

## **10.2.2** Task and computational model

We propose to employ an online physical effort for reward task to mimic decisions and behavior of effort and reward.

**Task:** The task is illustrated in Figure 5. Participants perform the task online at home on their computer, or they can also perform it in the lab on a computer. On each trial, patients need to decide between investing little effort (few button presses) for a small reward or more effort (more button presses) for a larger reward. Patients need to indicate their decision with the first button press within 4 sec and afterwards have 40 sec to execute their effortful behavior allowing to measure effort experience. On a subset of trials, participants are asked to rate their momentary happiness which we use as a proxy to assess reward experience. The task duration is around 25min. The task is written in javascript and can hence be run in any modern web browser. The data is saved on a GDPR-compliant cloud server within the EU (Google Firebase). Data will be pseudonymized throughout.

Analysis: To disentangle and quantify anticipation and experience separately for effort and reward we employ a generative computational model that captures the entire decision-making process. The model computes the values of a high effort/reward and a low effort/reward option including parameters relating to the effort and reward sensitivity implemented as a trade-off between necessary effort and the resulting reward (anticipation), the vigour used to execute the effortful behavior and the reaction to the reward (experience). The computed values are fed into a softmax function to determine the probability of making

a high effort/reward choice (Niv et al., 2007; Huys et al. 2013; Hauser et al., 2017; Berwian et al., 2020).

In our previous work (Berwian et al., 2020), we could show with the application of a computational model to the data collected by means of an earlier version of the task, that remitted, previously depressed, patients invested less effort for reward due to increased effort anticipation and that longer decision times prior to discontinuation (captured by larger boundaries in a drift-diffusion model) predicted later relapse better than chance in a validation sample. Hence, the task is established, could be used to disentangle effort anticipation and experience in a patient sample and provided robust effects. Based on our experience, we optimized the task as described above and established its validity by means of pilot data from healthy controls.

Analyses will be pre-registered. Moderation and mediation will be analyzed with linear mixed models with covariates x time x group interactions and mediation with dynamic panel models as outlined in the study protocol. Prediction will be examined using logistic regression in combination with an elastic net. The data will be split in advance into a training and validation sample.

You gained 7 points!
How happy does this reward make you?

1 point
20 button presses

1 point
20 button presses

1 point
20 button presses

1 point
20 button presses

Figure 5: Physical effort for reward task

### 10.2.3 Study design

The study design of the ChangePDD study is already established and depicted in Table 2. The additional task will be conducted at T1, T2, and T4 (V2, V5, and V11; see Table 2add-on). Data collected at T1 allows us to test hypothesis 1, while data collected at T2 and T4 allows us to assess hypothesis 2.

In addition, we will collect data with the task in matched healthy controls at T1 and T4. The healthy controls will be recruited in the context of the MAPPDD study. In the MaPPDD study,

144 healthy controls will be recruited using the infrastructure and funding already provided by the main study ChangePDD. Healthy controls will be recruited at the same six recruiting sites as the patients in ChangePDD. Each site will recruit 24 healthy controls, respectively. Screening will be performed to ensure that healthy controls are matched with patients regarding age and gender so that the healthy controls do not differ significantly from the PDD patients in the group comparison.

## 10.3. Study design and instruments supplemented by add-on studies

In order to get an overview of the design and the instruments when patients participate in both add-on studies in addition to ChangePDD, we have adapted Table 2 and Figure 3 accordingly.

**Table 2add-on:** Frequency and scope of trial visits of ChangePDD and the two add-on studies

| | Screening | | Inpat | ient I | | Inpatient II/Dayclinic | | | Conti | Continuationphase | | | Naturalistic follow-up | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Main Measurement Timepoints (T) | TO | T1 | | | T2 | inputient ii, bu | | T3 | Continuation | | T4 | Taranana raman ap | | | | | T5 |
| Trial Visits (V) | V1* | V2 | V3 | V4 | V5 | V6 | V7 | V8 | V9 | V10 | V11 | V12 | V13 | V14 | V15 | V16 | V17 |
| Week | pre | 1 | 2 | 4 | 5 | 6 | 8 | 10 | 12 | 14 | 16 | 24 | 32 | 40 | 48 | 56 | 64 |
| Informed Consent | X | | | | | | | | | - | - | - | | | | | |
| Random** | х | | | | | | | | | | | | | | | | |
| In-/Exclusion criteria | х | | | | | | | | | | | | | | | | |
| Patients master data | х | | | | | | | | | | | | | | | | |
| Patient preference | х | | | | | | | | | | | | | | | | |
| ATHF / concomitant medication | х | | | | | | | | | | | | | | | | |
| DIPS | х | | | | | | | | | | х | | | | | | х |
| SCID-5-PD | х | | | | | | | | | | х | | | | | | х |
| Primary Efficacy | | | | | | | | | | | | | | | | | |
| HDRS-24*** | х | х | | | х | | | х | | | Х | | | | | | x |
| Key secondary endpoints | | | | | | | | | | | | | | | | | |
| HDRS-24*** | х | х | х | х | | х | х | х | х | х | х | | | | | | х |
| IDS-SR | х | х | × | х | | x | x | × | х | х | х | х | х | х | х | х | x |
| BSI, GAF***, WHOQOL | х | х | | | х | | | х | | | х | | | | | | х |
| Response, remission, dropout-rate | | | | | х | | | х | | | х | | | | | | х |
| Relapse-rate | | | | | | | | | | | х | | | | | | х |
| Cost Interview | х | | | | | | | | | | х | | | | | | х |
| Further endpoints | | | | | | | | | | | | | | | | | |
| BDI-II, BRS, BSI, DAS, ECRRD8, ES, GSE,<br>IMI-R***, LQPT, MINI-ICF**, MPQ<br>PID5BF+M, RSQ, R-GPTS, SNI, UCLA,<br>WHOQOL, WBI | x | x | | | x | | | x | | | x | | | | | | x |
| Moderators of Change | | | | | | | | | | | | | | | | | |
| CTQ, BDNF methylation | х | | | | | | | | | | | | | | | | |
| Mediators of Change | | | | | | | | | | | | | | | | | |
| IIP-32-R, BADS, Step counts | x | х | x | х | | x | x | х | х | x | x | | | | | | x |
| Interpersonal Activation Diary**** | х | х | x | х | Х | x | | | | | | | | | | | |
| Social interaction and current mood | x | | | | | x | | | | | | | | | | | |
| Effort Task | | х | | | Х | | | | | | х | | | | | | |
| Side effects /( Serious) Adverse events | | | | | | | | | | | | | | | | | |
| SAEs and medication | | х | х | х | х | Х | Х | Х | х | Х | Х | | | | | | Х |
| SEPIPS | | | | | х | | | х | | | х | | | | | | х |
| Therapeutical Relationship, Adherence- | and Compete | nce Ra | ting, Sul | jective | Evalua | ion of Ir | mportan | t Doma | ins, The | rapist | | | | | | | |
| WAI, CBASP-CAR***, BA-CAR*** | | х | х | х | х | х | х | х | х | х | х | | | | | | |
| RevieW**** | | х | х х | х | х | х х | х х | х х | х х | х х | х х | | | | | | |
| THAT | | х | | | | | | | | | | | | | | | |

**Note.** Primary endpoint is marked red; \* V1 is divided into V1a to V1d (see Figure 3); \*\* Randomization will be performed between T0/V1 and T1/V2; \*\*\* Blinded observer ratings; \*\*\*\*In week pre and week 6, the IAD + (+ 2 items) will be used; \*\*\*\*\* Two crosses per cell because the questionnaire RevieW is done weekly

Figure 3add-on: Detailed Screening Flow supplemented by the two add-on studies



# 11. Safety

#### 11.1. Adverse reactions

**Adverse Event (AE)** is defined as any disadvantageous incident that occurs a person receiving either psychotherapeutic intervention, regardless of possible associations with the treatment received.

The following AES are defined for the study ChangePDD:

- Exacerbation of symptoms, e.g., generalization of symptoms
- Appearance of new symptoms
- Appearance of passive suicidal thoughts
- Appearance of active suicidal plans or intentions
- Occurrence of problems in the patient-therapist relation
- Further disadvantageous incidents as assessed by the therapist

**Adverse Treatment Reaction (ATR)** is defined as any AE due to a received treatment. The decision on the causality of AEs is made by the therapists and is supervised and controlled by the PI and Co-PIs and the DMC.

**Serious Adverse Events (SAE) and Serious Adverse Treatment Reactions (SATR)** are defined as an AE or ATR resulting in:

- Death
- Life-threatening event, e.g. suicidal attempt
- An incident requiring hospitalization

An incident leading to significant or permanent disability or invalidity.

(S)AEs and (S)ATRs are documented after each study treatment session (see 9.7 and 9.8) using an Adverse Event eCRF. In the eCRF, the corresponding therapist is asked to describe any adverse event, its duration (start/end date), intensity (mild, moderate, severe), assessment of causality (treatment related, probably related, unlikely related, not related, not assessable), the actions taken and the outcome of the action taken. In addition, the corresponding therapist is asked to assess whether the documented AEs and ATRs are judged serious (SAE, SATR).

In case of changing the individual therapists, the reasons for this change are documented in a separate form.

Adverse Event documentation is monitored during the study as part of the regulatory Monitoring conducted by the KKS Greifswald.

SAEs and SATRs must be reported electronically (via fax or e-mail) to the PI and the KKS Greifswald immediately within 24 hrs using a Serious Adverse Event report form that provides further details on the incident.

Patients who withdraw from study interventions due to one or more of the above mentioned reasons will be followed up in accordance with good clinical practice until a solution is found or the event is no longer considered clinically significant.

## 11.2. Risk-benefit-assessment

#### 11.2.1. Potential risks

As all patients are treatment-resistant and there is no placebo group, ethical concerns seem limited. Study participants will be treated with methods for which efficacy has been demonstrated in prior studies in severely depressed patients. The in/exclusion criteria were chosen to minimize the risks to patients.

However, in any psychotherapeutic treatment, there can be a temporary burden of actively dealing with topics discussed in the therapy sessions and possibly avoided so far. Under certain circumstances this can lead to the occurrence or increase of suicidal tendencies (suicidal thoughts or plans). Patients are regularly questioned on the subject of suicidal thoughts; in addition, they are asked to contact the study staff or appropriate emergency services at any time if they have suicidal thoughts.

Completing the questionnaires and conducting the interviews throughout the study (especially at the beginning) can also be potentially stressful for patients.

Patients are asked to immediately report any deterioration in their health status to the study staff, regardless of whether it is related to the scientific study. During the inpatient stay, patients can visit therapists from their treatment team at any time and during the dayclinic phase they can contact study staff (contact details are provided on the study information sheet). If stress becomes too great, patients can stop filling out questionnaires, conducting interviews or even participating in the entire study at any time without experiencing any disadvantages. If the study is discontinued, the patients will continue to be treated in the clinic as a 'non-study patient' according to the indication.

During the clinical trial, patients are also given a one-time blood sample (approx. 10 ml). The taking of a blood sample is usually associated with a very low risk. There may be slight pain at the puncture site or bruising, which may be visible for a few days. In extremely rare cases, a blood clot may form (thrombosis), a localised inflammation or infection may occur at the puncture site, or permanent damage to blood vessels or nerves may occur.

The DMC will monitor safety issues every 6 to 12 months. The informed consent process will be carefully conducted.

#### 11.2.2. Potential benefit

In this study, two psychotherapy programs (CBASP and BA) are examined with regard to their effectiveness in treating PDD with TR. It is known that both therapies have a positive influence on PDD. Whether one of the two therapies is better than the other in this indication is to be found out with this study. By participating, the study patients generally make a valuable scientific and health policy contribution to improving inpatient psychotherapy concepts in the short and long term.

The following concrete advantages and opportunities may also result from participation in the study for study-patients:

- Shortening of the waiting time until admission to the clinic
- Valuable and comprehensive diagnostics of the individual problems during the entire treatment
- An intensive psychotherapeutic inpatient and dayclinic depression treatment
- Participation in an outpatient group therapy after discharge to maintain the success and to prevent relapse
- Being part of a larger scientific study with close supervision by trained staff who are always available to patients

The overall results of this scientific study should contribute to finding an effective treatment for the group of PDD patients with treatment-resistance and increase the allocation of the patient to the individually more suitable therapy approach.

With regard to the health policy perspective, the following potential benefits should be pointed out: Considering the seriousness of the disease with its high risks for suicidality, low response to standard treatments as well as the enormous economic burden of an estimated 1 billion € annually in Germany, new evidence-based treatment programs are urgently needed to overcome TR and severely improve the current treatment of patients with PDD. The results provided by this study then have the potential to enable the establishment of the inpatient CBASP program in Germany (as well as other countries) and thereby vastly improving the current treatment of this serious disease.

#### 11.2.3. Conclusion

In view of the limited ethical concerns and potential risks mentioned and the continuous monitoring of safety issues, the overall potential risks in conducting the study appear to be low. Therefore, the described benefits of conducting the study, which have the potential to provide the results needed to significantly improve the current treatment of severe PDD with treatment-resistance, will outweigh the costs and potential risks.

#### 11.3. Discontinuation criteria

### 11.3.1. Premature discontinuation of a patient

In accordance with the Declaration of Helsinki, the patient's participation in the study is voluntary and each patient may withdraw from the study at any time without giving reasons for this decision. The decision to withdraw from the study treatment must be without any prejudice for the patient.

Study treatment of a patient may be terminated by the investigator for one or more of the following reasons:

- Active suicidality
- Physical health of the patient is a risk due to clinical judgement
- Occurrence of an AE/SAE (Averse Event/Serious Adverse Event) with therapeutic implications
- A newly emerging exclusion criterion
- Withdrawn of the informed consent
- Non-compliance with the study protocol

If the investigator terminates the treatment of the patient prematurely, he has to inform the patient about his decision and has to record the primary reason for withdrawal in the patient file and to document the end of treatment in the eCRF. If the patient caused the premature withdrawal the data collected before termination may be used if the patient agrees and an informed consent for follow up is signed by the patient.

#### 11.3.2. Premature discontinuation of the study

#### Single site

If a Leading Investigator has ethical concerns because of the performance at one of the sites, the Coordinating Investigator (PI) and the Co-PIs must be informed immediately.

The Coordinating Investigator together with the KKS Greifswald are authorized to discontinue this study at any time in any single site. Possible reasons for termination of the site could be but are not limited to:

- Unsatisfactory enrollment with respect to quantity or quality
- Inaccurate or incomplete data collection
- Unexpected accumulation of safety issues
- Major failure to adhere to the study protocol

### Study as a whole

The Coordinating Investigator together with the KKS Greifswald have the right to terminate this clinical study as a whole at any time. Possible reasons for termination of the study could be but are not limited to:

- Unexpected accumulation of safety issues
- Change of risk-benefit considerations

A premature discontinuation of a single site or of the study as a whole must be documented adequately with reasons being stated and information must be conveyed according to national requirements (e.g. Ethics Committee).

## 11.4. Data Monitoring Committee (DMC)

A Data Monitoring Commitee (DMC) has been established for this study consisting of one psychologist (Prof. Dr. Matthias Berking), one psychiatrist (Prof. Dr. Stefan Röpke), and one biostatistician (Prof. Dr. Michael Eid) – all highly experienced researchers in the field of clinical trials. The function of the DMC is to monitor the course and progress of the study against the predefined milestones and – if necessary – to give recommendations to the study administration for discontinuation, modification, or continuation of the study. The underlying principles for the DMC are ethical and safety aspects for the patients. It is the task of the DMC to examine whether the conducting of the study is still ethically justifiable, whether security of the patients is ensured, and whether the process of the study is acceptable. For this, the DMC is informed about the adherence to the protocol, patient recruitment, and the observed adverse events. The DMC will meet three times: 1) 6 months after "first patient in", 2) 18 months after "first patient in" and 3) 30 months after "first patient in", which should correspond to "last patient in" according to the study plan.

The outcome of the meetings is communicated to the Trial Steering Committee and the Leading Investigators of each site so that any administrative action required can be implemented.

In addition, Prof. Dr. Pim Cuijpers, Prof. Dr. Giovanni Fava, and Prof. Dr. Martin Hautzinger constitute the international Scientific Advisory Board (SAB). Due to their excellent expertise in conducting and analyzing clinical trials, they have been invited for providing independent advice and consulting regarding scientific, ethical, and data security issues, the dissemination process and external developments that are relevant to the progress and impact of the project.

## 12. Ethical and regulatory aspects

### 12.1. Laws and regulations

Good Clinical Practice (GCP) is an international ethical and scientific quality standard for designing, conducting, recording, and reporting studies that involve the participation of human patients. The study will be conducted in compliance with the guidelines of GCP and the applicable national laws and regulations (Berufsordnung der Ärzte und Psychotherapeuten) to assure that the rights, safety, and well-being of the participating patients are protected consistent with the ethical principles that have their origin in the Declaration of Helsinki.

## 12.2. Independent ethics committee

The study will only be started after consultation with the responsible ethics committee and only if there are no ethical concerns. The principal investigator (Prof. Dr. Brakemeier) is responsible for submitting the application to the Ethics Committee.

## 12.3. Changes to the study protocol

After the commencement of the clinical study, the Coordinating Investigator may amend the

protocol. If those amendments are substantial and are likely to have an impact on the safety of the study patients or to change the interpretation of the scientific documents in support of the conduct of the study, or if they are otherwise significant, the Coordinating Investigator shall notify the involved ethics committees.

If the opinion of the Ethics Committee is favourable the Coordinating Investigator shall proceed to conduct the clinical study following the amended protocol.

Amendments will be signed by all signatories of the protocol. All investigators will acknowledge the receipt and confirm by their signature on the amendment that they will adhere to the amendment. A copy of the signature page will be filed in the Investigator Study the original will be filed in the Trial Master File.

#### 12.4. Informed consent and insurance

A patient can only be included to the study if he/she has given his/her consent. A physician/therapist has to inform the patient verbally and in written form about the nature, meaning and scope of the study in an appropriate and understandable manner. The patient must have had sufficient time to make the decision. At the same time, with the consent, he/she must have declared that he/she agreed to the data being recorded as part of the study. The patient is informed that he/she can withdraw his/her consent at any time and without giving reasons without incurring disadvantages. If new information emerges during the course of the study that could influence the patient's willingness to participate, the Informed Consent Form will be changed accordingly. The patient is informed of the changes by a physician/therapist. Subsequently (assuming sufficient time to consider), the consent of the investigating physician/therapist and the patient must be signed again. An original of the patient's written information and consent is given to the patient. A second original is kept safe at the study site in the Investigator Site File (ISF).

During the study, no additional invasive or stressful examinations are carried out. The course of the study corresponds to the clinical routine. There are no study-related risks for the patient. Accordingly, it is not planned to take out subject insurance. An accident insurance is taken out for all patients for their dayclinic visits and the subsequent follow-up visits.

### 12.5. Data safety

The provisions of the data protection laws (EU-DSGVO) are observed. It is ensured that all examination data are pseudonymized adequately in accordance with the data protection regulations before scientific exploitation. An assignment of the personal data to the study data is only possible by the locally responsible study physician/therapist.

The study management (Prof. Dr. Eva-Lotta Brakemeier) receives the pseudonymized study data only for the purpose of scientifically evaluating the observational study. Exceptions to this are the video-based data of psychotherapies, which are used as described for supervision purposes, the CAR Ratings and research (concerning psychotherapy and depression research).

## 13. Statistics

## 13.1. Sample size

### **Analysis populations**

The Intent-to-treat (ITT) population will be defined as all patients randomized, regardless of whether they actually received treatment.

The Per Protocol (PP) population will be a subgroup of the ITT population that includes all patients who have been included in the trial, have no major protocol violation and who have participated in at least 16 individual sessions and 16 group therapies.

## Safety population

The safety population will be defined as all patients randomized who received at least one session of CBASP or BA.

## Sample size

Power calculation was based on a simulation study as recommended for linear-mixed effects models (Gelman & Hill, 2007). We intended the sample size to be large enough so that the power to detect a difference in the changes between treatments (CBASP vs. BA) of at least 3 HDRS points after 16 weeks is roughly 90% (assuming alpha = .05). This target effect size is in line with the NICE guidelines (Middleton et al., 2005), stating that a difference between groups of at least three points on the HDRS (and only two points for depression with TR) is clinically relevant. This also corresponds to Schramm et al. (2017) reporting a significant difference between CBASP and nonspecific psychotherapy of 2.5 on the HDRS after 20 weeks of outpatient-treatment (d = 0.31). Notably, this criterion is also supported by our CBASP metaanalysis that showed a significant combined overall effect size of small to moderate magnitude of CBASP versus other treatments or treatment as usual (TAU) (g = 0.34-0.44) (Negt et al., 2016). For the simulation study, Schramm et al. (2017) has been followed, in defining time as log transformed weeks after treatment onset and set the target treatment x time interaction effect to y = 1.06 (=3/log(16+1)). The remaining parameter values (e.g., random variances and covariance) were selected according to the results of Schramm et al. (2017), who shared their original HDRS data with us. Given these parameter values, the expected standard deviation of HRDS scores after 16 weeks is SD = 8.85, and thus the target effect of three HRDS points corresponds to a standardized effect of d = 0.34. Moreover, it is assumed that each person is assessed four times across the 16 weeks interval. A 14% dropout at primary endpoint is expected (assuming a linear increase of missing data across time). Given these parameters, the simulation (performed with the statistical platform R using 2000 resamples) suggests that a total sample size of N = 396 yields a power of 90% to detect the target interaction effect. Note that this estimate already takes into account that we expect about 14% missing data at the primary endpoint (i.e., after 16 weeks). Simulations including effects of covariates (e.g., recruitment sites) result in virtually identical estimates.

#### 13.2. Statistical evaluation

### 13.2.1. Primary endpoint

Differences in HDRS-24 change between experimental (CBASP) and control (BA) group will be analyzed using a linear mixed-effects model (LMM). In particular, the HDRS-24 scores across the 16 weeks will be predicted from log transformed time (i.e., weeks after treatment onset), treatment group, and their interaction. To account for unexplained individual differences in baseline status and rate of change, (correlated) random coefficients for the intercept and slope will be included. A p value <0.05 is considered to be significant. To consider the influence of strata (depression severity and participating site) and possible confounders (e.g., age, gender), the effect of respective baseline values will be explored (including interaction effects with time and treatment group). The primary analysis will be conducted in the intention-to treat (ITT) population using maximum likelihood estimation (ML) taking into account all available data points. ML yields accurate parameter estimates if values are missing at random

(MAR; i.e., values are missing at random conditional on other information in the model). Sensitivity analyses (including pattern mixture models; Hedeker & Gibbons, 1997) will be conducted to test whether the assumption that values are MAR is tenable. In case that missingness depends on other observed variables not included in the statistical model, a multilevel multiple imputation approach will be used (Enders et al., 2016). In case of nonnormally distributed residuals or heteroscedasticity, robust standard errors or, if appropriate, robust LMM will be used (Koller, 2016). Additionally, a per protocol analysis will be conducted to compare the results with the ITT population. Other details of the statistical analysis will be fixed in the Statistical Analysis Plan, to be prepared before start of the study (first patient in). All statistical analysis will be done with the software R (current version: 3.6.3) and Mplus (current version: 8.4).

### 13.2.2. Secondary endpoints

Secondary endpoints will also be analyzed with (generalized) LMM. Moderator variables will be evaluated within these models by including interaction effects of moderator baseline values with time and treatment group. Mediator variables will be evaluated using dynamic panel models (Falkenström et al., 2017).

### 13.2.3. Safety and tolerability endpoints

Safety analyses will be performed for all patients having started one of the treatments. Patients will be analyzed according to treatment received. Rates of adverse events and SAEs will be calculated with corresponding two-sided 95% confidence intervals.

### 13.2.4. Handling of dropouts

It is expected that 5% of the patients will drop out of the study directly after the randomization, and further 10% will drop out during treatment. Therefore, we expect 95% x 90% = 85.5% of randomized patients to have HDRS-24 non-missing in week 16. All available data points will be used to estimate model parameters using maximum likelihood estimation. Thus, we will include earlier data points from patients who drop out of the study as long as they do not withdraw consent. Moreover, all efforts will be made during the informed consent procedure to include only patients who are willing to accept both arms and to continue study visits until W64/T5 irrespectively of compliance.

The dropout patients receive the standard treatment of the corresponding ward, so that clinically there are no disadvantages for the patients due to a dropout.

### 14. Data Management

### 14.1. Data collection

All data on patients collected in eCRFs and CRFs during the course of the study will be documented pseudonymously, i.e. the patient will be identified only by the pseudonymized identification number. Investigator must ensure that the patient's encryption is maintained. The patient identification list should be kept in strict confidence at the study site in the ISF. The investigator at each study site is responsible for keeping the identification list and informed consent forms locked up.

Most of the information required by the protocol and collected during the trial is entered directly into the eCRF electronically by patients or by the investigators or a designated representative. Some information required under the protocol that cannot be entered directly

into the eCRF electronically is entered into the CRF by the investigators or a designated representative.

The investigator will maintain a list of individuals authorized to enter or correct data (study delegation log).

## 14.2. Data processing

## 14.2.1 EDC-System (eCRF)

The data of the patients are documented within the EDC (Electronic Data Capture) system eHealth-Platform. Data will be entered by study personnel as well as directly by patients. The data of the actimeter are read from the clock during the bi-weekly study visit and entered into the eCRF by the study personnel (rater). Data are entered directly via web browser to the eCRF. Detailed instructions for using the EDC system are specified in the EDC Manual, which is part of the ISF.

In order to use the EDC system all staff who are entering and monitoring data are provided with training materials and required documentation by the KKS Greifswald. All data which are collected during the trial have to be documented in the eCRF by authorized persons according to the Delegation log. Specific user roles within the system enforce accordance with the Delegation Log.

The EDC system has an implemented audit trail. This assures that any documentation and/or changes to database items are traceable anytime. Changes or corrections are permitted to authorized persons who have access to the system with user specific access rights. This access is documented in the audit trail. Users with monitoring function are not able to enter or change patient's data. They have the possibility to view the data write protected (review function) and they can create SDV marks in case of queries. Discrepancies which appear at data management are forwarded to the monitors or to the site directly.

#### 14.2.2 Data concealment for electronic transfer

The eHealth-Platform uses personalized certificate to ensure authorized access. Stored data are further secured with regular backups. At the end of study, the database will be closed after data cleaning process.

### **14.2.3** Data discrepancies

In a multistage procedure, the obtained data will be checked electronically for their plausibility and consistency. Detected inconsistencies and missing or implausible data will be clarified with queries and necessary changes will be carried out.

#### 14.2.4 Registration

Before recruitment and data collection starts, the trial will be registered at Clinical trials (http://clinicaltrials.gov) and DRKS (<a href="www.germanctr.de">www.germanctr.de</a>). Prof. Dr. Eva-Lotta Brakemeier is responsible for the first registration and following updates.

#### 14.2.5 Publication

The study results are presented at scientific symposia and published in international journals according to the criteria of the CONSORT declaration, regardless of the result. At least within one year after completion of the study, the main manuscript will be completed for publication. Any formal presentation or publication of data collected as a direct or indirect result of this study will be considered by the investigators as a joint publication. It therefore requires the agreement of the Coordinating Investigator and the Co-Principal Investigators. The authorship will be determined by mutual agreement.

The results of this study may be presented at scientific symposia or published in a scientific journal only after review and written approval by the Coordinating Investigator and the Co-Principal Investigators. The Investigators of the participating centers agree not to make presentations based on data collected individually or from a subset of centers prior to the publication of the first main publication, unless otherwise agreed by all other investigators, the Coordinating Investigator, and the Co-Principal Investigators.

The Coordinating Investigator, the Co-Principle Investigators and all Leading Investigators will receive copies of all communications, presentations or publications within a reasonable time in advance (at least 10 working days for an abstract or oral presentation material and 35 working days for a manuscript). These guidelines are provided to check the communications for accuracy, to ensure that confidential information is not inadvertently disclosed, to allow for appropriate input or additional information that may not have been available to the Investigator, and to allow for co-authorship.

#### 14.2.6 Open Data

In accordance with the Open Science specifications of the German Psychological Association (DGPs), anonymized data is made available to the public via the Open Data portal of the Open Science Foundation (ww.osf.io). The data will be stored when data collection is completed, but not before 01.01.2028. This step allows third parties to reproduce the analyses reported in scientific publications and to perform ad hoc analyses. The data is permanently stored on servers located in Germany. As soon as they are uploaded and published, these anonymized data cannot be deleted and are therefore also excluded from the deletion of the data in case of revocation of the study participation.

## 14.3. Quality assurance and quality control

#### 14.3.1. Source data and subject files

The investigator has to keep a written or electronic subject/patient file for every subject participating in the clinical study. In this file, the available demographic and medical information of a subject has to be documented, in particular the following: name, date of birth, sex, height, weight, subject history, concomitant diseases and concomitant drug (including changes during the study), statement of entry into the study, study identification, subject number, the date and process of informed consent, all study visit dates, predefined performed examinations and clinical findings, observed (S)AEs (if applicable), and reason for withdrawal from the study if applicable. It must be possible to identify each subject by using this patient file.

Additionally, any other documents with source data, especially original printouts of data that were generated by technical equipment have to be filed. All these documents have to bear at least subject identification and the printing date printed by the recording device to indicate to which subject and to which study procedure the document belongs. The medical evaluation of such records should be documented as necessary and signed/dated by the investigator.

For the current study, documents considered to be source data include (but are not limited to):

- Patient's record (patient's clinic and/or office chart, hospital chart).
- Patient Informed Consent Form
- Laboratory results
- Pharmacy records
- Treatment notes
- Scores
- Any other records maintained to conduct and evaluate the clinical study

#### 14.3.2. Monitoring

During the course of the study each participating site will be visited for monitoring before, during and after the study. During each of these visits, source data verification will be performed based on the monitoring plan, generated by the KKS Greifswald. The monitoring of the study takes place by the trained staff of the KKS Greifswald. Content, amount and details of the monitoring visits are described in the monitoring plan. Additionally, on-site and remotemonitoring visits are defined.

In general, any discrepancies in the data collection should be discussed and clarified with the study team during the monitoring visit and corrections/additions should be done according to GCP requirements.

All Monitoring visits are documented according to KKS-specific SOPs.

#### 15. Literature

Angermeyer, M. C., Kilian, R., & Matschinger, H. (2000). WHOQOL-100 und WHOQOL-BREF. Handbuch für die deutschprachige Version der WHO Instrumente zur Erfassung von Lebensqualität. Hogrefe.

Angst, J., Gamma, A., Rössler, W., Ajdacic, V., & Klein, D. N. (2009). Long-term depression versus episodic major depression: Results from the prospective Zurich study of a community sample. *Journal of Affective Disorders*, *115*(1–2), 112–121. <a href="https://doi.org/10.1016/j.jad.2008.09.023">https://doi.org/10.1016/j.jad.2008.09.023</a>

Asparouhov, T., Hamaker, E. L., & Muthén, B. (2018). Dynamic Structural Equation Models. Structural Equation Modeling: A Multidisciplinary Journal, 25(3), 359–388. https://doi.org/10.1080/10705511.2017.1406803

Association, A. P. *Diagnostic and Statistical Manual of Mental Disorders (DSM-5®)*. (American Psychiatric Pub, 2013).

Bach, B., Kerber, A., Aluja, A., Bastiaens, T., Keeley, J. W., Claes, L., Fossati, A., Gutierrez, F., Oliveira, S. E. S., Pires, R., Riegel, K. D., Rolland, J.-P., Roskam, I., Sellbom, M., Somma, A., Spanemberg, L., Strus, W., Thimm, J. C., Wright, A. G. C., & Zimmermann, J. (in press). International assessment of DSM-5 and ICD-11 personality disorder traits: Toward a common nosology in DSM-5.1. *Psychopathology*. <a href="https://doi.org/10.1159/000507589">https://doi.org/10.1159/000507589</a>

- Bajbouj, M., Aust, S., Spies, J., Herrera-Melendez, A.-L., Mayer, S. V., Peters, M., Plewnia, C., Fallgatter, A. J., Frase, L., Normann, C., Behler, N., Wulf, L., Brakemeier, E.-L., & Padberg, F. (2018). PsychotherapyPlus: Augmentation of cognitive behavioral therapy (CBT) with prefrontal transcranial direct current stimulation (tDCS) in major depressive disorder—study design and methodology of a multicenter double-blind randomized placebocontrolled trial. *European Archives of Psychiatry and Clinical Neuroscience*, 268(8), 797—808. <a href="https://doi.org/10.1007/s00406-017-0859-x">https://doi.org/10.1007/s00406-017-0859-x</a>
- Beesdo-Baum, K., Zaudig, M., Wittchen, H.-U., (2019). Strukturiertes Klinisches Interview für DSM-5-Persönlichkeitsstörungen. Deutsche Bearbeitung des Structured Clinical Interview for DSM-5 Personality Disorders von Michael B. First, Janet B.W. Williams, Lorna Smith Benjamin, Robert L. Spitzer. Hogrefe.
- Bernstein, D.P., Stein, J.A., Newcomb, M.D., Walker, E., Pogge, D., Ahluvalia, T., Stokes, J., Handelsman, L., Medrano, M., Desmond, D., Zule, W., 2003. Development and validation of a brief screening version of the Childhood Trauma Questionnaire. *Child Abuse & Neglect*, *27*, 169–190. <a href="https://doi.org/10.1016/S0145-2134(02)00541-0">https://doi.org/10.1016/S0145-2134(02)00541-0</a>
- Berwian, I. M., Wenzel, J., Collins, A.G.E., Seifritz, E., Stephan, K.E., Walter, H., Huys, Q.J.M., 2020. Computational mechanisms of effort and reward decisions in patients with depression and their association with relapse after antidepressant discontinuation. *JAMA psychiatry*. https://doi.org/10.1001/jamapsychiatry.2019.4971
- Brakemeier, E.-L., Dobias, J., Hertel, J., Bohus, M., Limberger, M. F., Schramm, E., Radtke, M., Frank, P., Padberg, F., Sabass, L., Jobst, A., Jacob, G. A., Struck, N., Zimmermann, J., & Normann, C. (2018). Childhood Maltreatment in Women with Borderline Personality Disorder, Chronic Depression, and Episodic Depression, and in Healthy Controls. *Psychotherapy and Psychosomatics*, *87*(1), 49–51. <a href="https://doi.org/10.1159/000484481">https://doi.org/10.1159/000484481</a>
- Brakemeier, E.-L., Engel, V., Schramm, E., Zobel, I., Schmidt, T., Hautzinger, M., Berger, M., & Normann, C. (2011). Feasibility and Outcome of Cognitive Behavioral Analysis System of Psychotherapy (CBASP) for Chronically Depressed Inpatients: A Pilot Study. *Psychotherapy and Psychosomatics*, 80(3), 191–194. <a href="https://doi.org/10.1159/000320779">https://doi.org/10.1159/000320779</a>
- Brakemeier, E.-L., Herzog, P., Radtke, M., Schneibel, R., Breger, V., Becker, M., Spies, J., Jacobi, F., Heider, J., & Normann, C. (2018). CBASP als stationäres Behandlungskonzept der therapieresistenten chronischen Depression: Eine Pilotstudie zum Zusammenhang von Nebenwirkungen und Therapieerfolg. *PPmP Psychotherapie · Psychosomatik · Medizinische Psychologie*, 68(09/10), 399–407. https://doi.org/10.1055/a-0629-7802
- Brakemeier, E.-L., Marchner, J., Gutgsell, S., Engel, V., Radtke, M., Tuschen-Caffier, B., Normann, C., & Berking, M. (2013). CBASP@home: Ein internetbasiertes Situationsanalysen-Training zur Stabilisierung des Therapieerfolgs nach stationärer Therapie für chronisch depressive Patienten. *Verhaltenstherapie*, *23*(3), 190–203. <a href="https://doi.org/10.1159/000354814">https://doi.org/10.1159/000354814</a>
- Brakemeier, E.-L., Merkl, A., Wilbertz, G., Quante, A., Regen, F., Bührsch, N., & Kathmann, N. (2014). Continuation treatment after electroconvulsive therapy in patients with unipolar depression. *Biological Psychology*, *76*, 194–202. https://doi.org/10.1016/j.biopsych.2013.11.030
- Brakemeier, E.-L., & Normann, C. (2012). *Praxisbuch CBASP: Behandlung chronischer Depression; mit Online-Materialien* (1. Aufl). Beltz.
- Brakemeier, E.-L., Guhn, A., & Normann, C. (in press). *Praxisbuch CBASP: Behandlung chronischer Depression und Modifikationen für weitere interpersonelle Störungen; mit E-Book inside und Arbeitsmaterial;* (2., überarbeitete und erweiterte Auflage). Beltz.

- Brakemeier, E.-L., Radtke, M., Engel, V., Zimmermann, J., Tuschen-Caffier, B., Hautzinger, M., Schramm, E., Berger, M., & Normann, C. (2015). Overcoming Treatment Resistance in Chronic Depression: A Pilot Study on Outcome and Feasibility of the Cognitive Behavioral Analysis System of Psychotherapy as an Inpatient Treatment Program. *Psychotherapy and Psychosomatics*, 84(1), 51–56. <a href="https://doi.org/10.1159/000369586">https://doi.org/10.1159/000369586</a>
- Bschor, T., Bauer, M., & Adli, M. (2014). Chronic and Treatment Resistant Depression. *Deutsches Aerzteblatt Online, 111,* 766-776. https://doi.org/10.3238/arztebl.2014.0766
- Buecker, S., Horstmann, K. T., Terwiel, S., Krasko, J., Kritzler, S., Kaiser, T., & Luhmann, M. (2020, June 3). Psychological Item Pool for Corona Outbreak (PIPCO). Retrieved from osf.io/62dmf
- Casper, F., Fingerle, H., & Werner, M. (2000). Der IMI (Impact Message Inventory): Ein Instrument zur interpersonalen Fremdbeurteilung. *Forschungsbericht aus dem psychologischen Institut der Universität Freiburg*. Thieme.
- Carrozzino, D., Patierno, C., Fava, G.A., & Guidi, J. (2020). The Hamilton Rating Scales for Depression: A Critical Review of Clinimetric Properties of Different Versions. *Psychotherapy and Psychosom*atics, 89(3), 133–150. https://doi:10.1159/000506879
- Carrozzino, D., Svicher, A., Patierno, C., Berrocal, C., & Cosci, F. (2019). The Euthymia Scale: A Clinimetric Analysis. *Psychotherapy and Psychosom*atics, 88(2), 119–121. https://doi:10.1159/000496230
- Chaix, R., Alvarez-López, M. J., Fagny, M., Lemee, L., Regnault, B., Davidson, R. J., Lutz, A., & Kaliman, P. (2017). Epigenetic clock analysis in long-term meditators. *Psychoneuroendocrinology*, 85, 210–214. <a href="https://doi.org/10.1016/j.psyneuen.2017.08.016">https://doi.org/10.1016/j.psyneuen.2017.08.016</a>
- Cohen, S., Doyle, W. J., Skoner, D. P., Rabin, B. S., & Gwaltney, J. M. (1997). Social ties and susceptibility to the common cold. *Jama*, *277*(24), 1940–1944. https://doi.org/10.1001/jama.1997.03540480040036
- Constantino, M. J., Manber, R., DeGeorge, J., McBride, C., Ravitz, P., Zuroff, D. C., Klein, D. N., Markowitz, J. C., Rothbaum, B. O., Thase, M. E., & Arnow, B. A. (2008). Interpersonal styles of chronically depressed outpatients: Profiles and therapeutic change. *Psychotherapy: Theory, Research, Practice, Training*, *45*(4), 491–506. https://doi.org/10.1037/a0014335
- Cuijpers, P., Clignet, F., van Meijel, B., van Straten, A., Li, J., & Andersson, G. (2011). Psychological treatment of depression in inpatients: A systematic review and meta-analysis. *Clinical Psychology Review*, *31*(3), 353–360. https://doi.org/10.1016/j.cpr.2011.01.002
- Cuijpers, P., van Straten, A., Schuurmans, J., van Oppen, P., Hollon, S. D., & Andersson, G. (2010). Psychotherapy for chronic major depression and dysthymia: A meta-analysis. *Clinical Psychology Review*, *30*(1), 51–62. https://doi.org/10.1016/j.cpr.2009.09.003
- Cuijpers, P., van Straten, A., & Warmerdam, L. (2007). Behavioral activation treatments of depression: A meta-analysis. *Clinical Psychology Review*, *27*(3), 318–326. https://doi.org/10.1016/j.cpr.2006.11.001
- Derogatis, L. R., & Spencer, P. M. (1993). *Brief symptom inventory: BSI*. Pearson, Upper Saddle River, NJ.
- DGPPN, BÄK, KBV, AWMF (2015). S3-Leitlinie/Nationale Versorgungsleitlinie Unipolare Depression- Langfassung: Bd. Version 5 (2. Aufl.). Springer.

- Dimidjian, S., Hollon, S. D., Dobson, K. S., Schmaling, K. B., Kohlenberg, R. J., Addis, M. E., Gallop, R., McGlinchey, J. B., Markley, D. K., Gollan, J. K., Atkins, D. C., Dunner, D. L., & Jacobson, N. S. (2006). Randomized trial of behavioral activation, cognitive therapy, and antidepressant medication in the acute treatment of adults with major depression. *Journal of Consulting and Clinical Psychology*, *74*(4), 658–670. https://doi.org/10.1037/0022-006X.74.4.658
- Döring, N., & Bortz, J. (1993). Psychometrische Einsamkeitsforschung: Deutsche Neukonstruktion der UCLA Loneliness Scale. *Diagnostica*, *39*, 224–239.
- Downey, G., & Feldman, S. I. (1996). Implications of rejection sensitivity for intimate relationships. *Journal of personality and social psychology*, *70* (6), 1327. https://doi.org/10.1037/0022-3514.70.6.1327
- Drummond, M. F. (Hrsg.). (2007). *Methods for the economic evaluation of health care programmes* (3. Aufl.). Oxford University Press.
- Ekers, D., Richards, D., & Gilbody, S. (2008). A meta-analysis of randomized trials of behavioural treatment of depression. *Psychological Medicine*, *38*(5), 611–623. https://doi.org/10.1017/S0033291707001614
- Enders, C. K., Mistler, S. A., & Keller, B. T. (2016). Multilevel multiple imputation: A review and evaluation of joint modeling and chained equations imputation. *Psychological Methods*, *21*(2), 222–240. <a href="https://doi.org/10.1037/met0000063">https://doi.org/10.1037/met0000063</a>
- Fava, G.A., Tomba, E., Brakemeier, E.-L., et al. (2019). Mental Pain as a Transdiagnostic Patient-Reported Outcome Measure. *Psychotherapy and Psychosomatics*, *88*(6), 341–349. https://doi:10.1159/000504024
- Falkenström, F., Finkel, S., Sandell, R., Rubel, J. A., & Holmqvist, R. (2017). Dynamic models of individual change in psychotherapy process research. *Journal of Consulting and Clinical Psychology*, 85(6), 537–549. <a href="https://doi.org/10.1037/ccp0000203">https://doi.org/10.1037/ccp0000203</a>
- Forbes, C. N. (2020). New directions in behavioral activation: Using findings from basic science and translational neuroscience to inform the exploration of potential mechanisms of change [published online ahead of print, 2020 May 5]. *Clinical Psychology Review*, 79, 101860. <a href="https://doi:10.1016/j.cpr.2020.101860">https://doi:10.1016/j.cpr.2020.101860</a>
- Freeman, D. *et al.* (2019). The revised Green et al., Paranoid Thoughts Scale (R-GPTS): psychometric properties, severity ranges, and clinical cut-offs. *Psychological Medicine*, 1–10. https://doi.org/10.1017/S0033291719003155
- Frieling, H., & Tadić, A. (2013). Value of genetic and epigenetic testing as biomarkers of response to antidepressant treatment. *International Review of Psychiatry*, 25(5), 572–578. https://doi.org/10.3109/09540261.2013.816657
- Gelman, A., & Hill, J. (2007). *Data analysis using regression and multilevel/hierarchical models*. Cambridge University Press.
- Geyer, E.C., Fua, K.C., Daniel, K.E., Chow, P.I., Bonelli, W., Huang, Y., Barnes, L.E., and Teachman, B.A. (2018). I Did OK, but Did I Like It? Using Ecological Momentary Assessment to Examine Perceptions of Social Interactions Associated With Severity of Social Anxiety and Depression. *Behav Ther* 49, 866-880. <a href="https://doi.org/10.1016/j.beth.2018.07.009">https://doi.org/10.1016/j.beth.2018.07.009</a>
- Guhn, A., Köhler, S., Brakemeier, E.-L., & Sterzer, P. (2019). Cognitive Behavioral Analysis System of Psychotherapy for inpatients with persistent depressive disorder: a naturalistic trial on a general acute psychiatric unit. *European Archives of Psychiatry and Clinical Neuroscience*. 2019 Jul 12. https://doi.org/10.1007/s00406-019-01038-5

- Hall, R. C. W. (1995). Global Assessment of Functioning. *Psychosomatics*, *36*(3), 267–275. https://doi.org/10.1016/S0033-3182(95)71666-8
- Hamilton, M. (1960). A Rating Scale for Depression. *Journal of Neurology, Neurosurgery & Psychiatry*, 23(1), 56–62. <a href="https://doi.org/10.1136/jnnp.23.1.56">https://doi.org/10.1136/jnnp.23.1.56</a>
- Hauser, T.U. et al. Separate mesocortical and mesolimbic pathways encode effort and reward learning signals. *Proc Natl Acad Sci USA* (2017). https://doi.org/10.1073/pnas.1705643114
- Hautzinger, M., Joormann, J., & Keller, F. (2005). *DAS: Skala dysfunktionaler Einstellungen; Manual*. Hogrefe.
- Hautzinger, M., Keller, F., & Kühner, C. (2006). Das Beck Depressionsinventar II. Hogrefe.
- Hedeker, D., & Gibbons, R. D. (1997). Application of random-effects pattern-mixture models for missing data in longitudinal studies. *Psychological Methods*, *2*(1), 64–78. <a href="https://doi.org/10.1037/1082-989X.2.1.64">https://doi.org/10.1037/1082-989X.2.1.64</a>
- Herzog, P., Kaiser, T., Gärtner, T., Rief, W., & Brakemeier, E.-L. (in prep). Detecting and monitoring side effects of psychological interventions: Development and Validation of the Side Effects of Psychological Interventions Process Scale (SEPIPS)
- Hopko, D. R., Lejuez, C. W., Lepage, J. P., Hopko, S. D., & McNeil, D. W. (2003). A Brief Behavioral Activation Treatment for Depression: A Randomized Pilot Trial within an Inpatient Psychiatric Hospital. *Behavior Modification*, *27*(4), 458–469. https://doi.org/10.1177/0145445503255489
- Horowitz, L. M., Alden, L. E., Kordy, H., & Strauß, B. (2000). *Inventar zur Erfassung interpersonaler Probleme: Deutsche Version; IIP-D.* Beltz.
- Hörter, M., Sitta, P., Keller, F., Metzger, R., Wiegand, W., Schell, G., Stieglitz, R.-D., Wolfersdorf, M., Felsenstein, M., & Berger, M. (2004). Stationäre psychiatrisch-psychotherapeutische Depressionsbehandlung: Prozess- und Ergebnisqualität anhand eines Modellprojekts in Baden-Württemberg. *Der Nervenarzt*, 75(11), 1083–1091. https://doi.org/10.1007/s00115-004-1705-8
- Hölzel, L., Wolff, A. von, Kriston, L., & Härter, M. (2010). Unter welchen Bedingungen bleibt eine stationäre Depressionsbehandlung erfolglos? *Psychiatrische Praxis*, *37*(01), 27–33. https://doi.org/10.1055/s-0029-1223348
- Huys, Q.J.M. et al. Mapping anhedonia onto reinforcement learning: a behavioural metaanalysis. *Biol Mood Anxiety Disord* (2013). https://doi.org/10.1186/2045-5380-3-12
- Jacobs, I., & Scholl, W. (2005). Interpersonale Adjektivliste (IAL). *Diagnostica*, *51*(3), 145–155. <a href="https://doi.org/10.1026/0012-1924.51.3.145">https://doi.org/10.1026/0012-1924.51.3.145</a>
- Jacobs, I., & Scholl, W. (2016). IAL-K: Entwicklung einer Kurzform der Interpersonalen Adjektivliste. *Diagnostica*, 62(4), 227–241. https://doi.org/10.1026/0012-1924/a000156
- Jobst, A., Brakemeier, E.-L., Buchheim, A., Caspar, F., Cuijpers, P., Ebmeier, K. P., Falkai, P., Jan van der Gaag, R., Gaebel, W., Herpertz, S., Kurimay, T., Sabaß, L., Schnell, K., Schramm, E., Torrent, C., Wasserman, D., Wiersma, J., & Padberg, F. (2016). European Psychiatric Association Guidance on psychotherapy in chronic depression across Europe. *European Psychiatry*, *33*, 18–36. <a href="https://doi.org/10.1016/j.eurpsy.2015.12.003">https://doi.org/10.1016/j.eurpsy.2015.12.003</a>
- Kahl, K. G., Winter, L., & Schweiger, U. (2012). The third wave of cognitive behavioural therapies: What is new and what is effective? *Current Opinion in Psychiatry*, *25*(6), 522–528. <a href="https://doi.org/10.1097/YCO.0b013e328358e531">https://doi.org/10.1097/YCO.0b013e328358e531</a>
- Kanter, J. W. (2009). *Behavioral Activation: Distinctive Features* (1. Aufl.). Routledge. https://doi.org/10.4324/9780203876060

- Kanter, J. W., Mulick, P. S., Busch, A. M., Berlin, K. S., & Martell, C. R. (2007). The Behavioral Activation for Depression Scale (BADS): Psychometric Properties and Factor Structure. *Journal of Psychopathology and Behavioral Assessment*, 29(3), 191–202. <a href="https://doi.org/10.1007/s10862-006-9038-5">https://doi.org/10.1007/s10862-006-9038-5</a>
- Keller, F., Härter, M., Metzger, R., Wiegand, W., & Schell, G. (2001). Prozess-und Ergebnisqualität in der stationären Behandlung ersterkrankter und chronisch depressiver Patienten. *Krankenhauspsychiatrie*, *12*(1), 50–56. <a href="http://dx.doi.org/10.1055/s-2001-17668">http://dx.doi.org/10.1055/s-2001-17668</a>
- Keller, Martin B., McCullough, J. P., Klein, D. N., Arnow, B., Dunner, D. L., Gelenberg, A. J., Markowitz, J. C., Nemeroff, C. B., Russell, J. M., Thase, M. E., Trivedi, M. H., Blalock, J. A., Borian, F. E., Jody, D. N., DeBattista, C., Koran, L. M., Schatzberg, A. F., Fawcett, J., Hirschfeld, R. M. A., ... & Zajecka, J. (2000). A Comparison of Nefazodone, the Cognitive Behavioral-Analysis System of Psychotherapy, and Their Combination for the Treatment of Chronic Depression. New England Journal of Medicine, 342(20), 1462–1470. <a href="https://doi.org/10.1056/NEJM200005183422001">https://doi.org/10.1056/NEJM200005183422001</a>
- Keller, M.B., Warshaw, M. G., Dyck, I., Dolan, R. T., Shea, M. Y., Riley, K., & Shapiro, R. (1997). LIFE-IV: The Longitudinal Interval Follow-up Evaluation for DSM-IV.
- Kerber, A., Schultze, M., Müller, S., Rühling, R. M., Wright, A. G., Spitzer, C., Krueger, R., ... & Zimmermann, J. (2019). *Development of a Short and ICD-11 Compatible Measure for DSM-5 Maladaptive Personality Traits Using Ant Colony Optimization Algorithms*. <a href="https://doi.org/10.31234/osf.io/rsw54">https://doi.org/10.31234/osf.io/rsw54</a>
- Klein, J. P., Erkens, N., Schweiger, U., Kriston, L., Bausch, P., Zobel, I., Hautzinger, M., Schoepf, D., Serbanescu, I., Bailer, J., Backenstrass, M., Wambach, K., Walter, H., Härter, M., & Schramm, E. (2018). Does Childhood Maltreatment Moderate the Effect of the Cognitive Behavioral Analysis System of Psychotherapy versus Supportive Psychotherapy in Persistent Depressive Disorder? *Psychotherapy and Psychosomatics*, 87(1), 46–48. <a href="https://doi.org/10.1159/000484412">https://doi.org/10.1159/000484412</a>
- Klug, G., Huber, D., & Kächele, H. (2002). *Psychotherapeutische Haltung (ThAt). Ein Fragebogen zur Ausbildung, Erfahrung, Stil und Werten*.
- Kocsis, J. H. (2009). Cognitive Behavioral Analysis System of Psychotherapy and Brief Supportive Psychotherapy for Augmentation of Antidepressant Nonresponse in Chronic Depression. The REVAMP Trial. *Archives of General Psychiatry*, 66(11), 1178. <a href="https://doi.org/10.1001/archgenpsychiatry.2009.144">https://doi.org/10.1001/archgenpsychiatry.2009.144</a>
- Köhler, S., Sterzer, P., Normann, C., Berger, M., & Brakemeier, E.-L. (2016). Überwindung der Therapieresistenz bei chronischer Depression: Die Bedeutung der stationären Psychotherapie. *Der Nervenarzt*, *87*(7), 701–707. <a href="https://doi.org/10.1007/s00115-015-0034-4">https://doi.org/10.1007/s00115-015-0034-4</a>
- Koller, M. (2016). robustlmm: An R Package for Robust Estimation of Linear Mixed-Effects Models. *Journal of Statistical Software*, 75(6). https://doi.org/10.18637/jss.v075.i06
- Koy, J. (2019). Specific and non-specific working mechanisms of inpatient psychotherapy concepts in patients with depression: Validation of the questionnaire "Review of last Week (RevieW). Masterthesis. Philipps-Universität Marburg.
- Krieger, T., Zimmermann, J., Huffziger, S., et al. (2014). Measuring depression with a well-being index: further evidence for the validity of the WHO Well-Being Index (WHO-5) as a measure of the severity of depression. *Journal of Affective Disorders*, 156, 240–244. <a href="https://doi.org/10.1016/j.jad.2013.12.015">https://doi.org/10.1016/j.jad.2013.12.015</a>

- Kriston, L., von Wolff, A., Westphal, A., Hölzel, L. P., & Härter, M. (2014). Efficacy and Acceptability of acute treatments for Persistent Depressive Disorder: A Network Meta-Analysis: Acute Treatments for Persistent Depressive Disorder. *Depression and Anxiety,* 31(8), 621–630. <a href="https://doi.org/10.1002/da.22236">https://doi.org/10.1002/da.22236</a>
- Köhler, S., Fischer, T., Brakemeier, E.-L., & Sterzer, P. (2015). Successful Treatment of Severe Persistent Depressive Disorder with a Sequential Approach: Electroconvulsive Therapy Followed by Cognitive Behavioural Analysis System of Psychotherapy. *Psychotherapy and Psychosomatics*, 84(2), 127–128. <a href="https://doi.org/10.1159/000369847">https://doi.org/10.1159/000369847</a>
- Köhler, S., Chrysanthou, S., Guhn, A., & Sterzer, P. (2019). Differences between chronic and nonchronic depression: Systematic review and implications for treatment. *Depression and Anxiety*, *36*(1), 18–30. <a href="https://doi.org/10.1002/da.22835">https://doi.org/10.1002/da.22835</a>
- Kühnen, T., Knappke, F., Otto, T., Friedrich, S., Klein, J., Kahl, K., Hüppe, M., Sipos, V. & Schweiger, U. (2011). Chronic depression: development and evaluation of the luebeck questionnaire for recording preoperational thinking (LQPT). *BMC Psychiatry*, *11*, 199. <a href="https://doi.org/10.1186/1471-244X-11-199">https://doi.org/10.1186/1471-244X-11-199</a>
- Lewinsohn, P. M. A behavioral approach to depression. *Essential papers on depression*, 150-172 (1974).
- Lieb, K., Dreimüller, N., Wagner, S., Schlicht, K., Falter, T., Neyazi, A., Müller-Engling, L., Bleich, S., Tadić, A., & Frieling, H. (2018). BDNF Plasma Levels and BDNF Exon IV Promoter Methylation as Predictors for Antidepressant Treatment Response. *Frontiers in Psychiatry*, *9*, 511. https://doi.org/10.3389/fpsyt.2018.00511
- Linden, M., & Baron, S. (2005). Das "Mini-ICF-Rating für psychische Störungen (Mini-ICF-P)". Ein Kurzinstrument zur Beurteilung von Fähigkeitsstörungen bei psychischen Erkrankungen. *Die Rehabilitation*, *44*(3), 144–151. <a href="https://doi.org/10.1055/s-2004-834786">https://doi.org/10.1055/s-2004-834786</a>
- Luborsky, L., Diguer, L., Seligman, D. A., Rosenthal, R., Krause, E. D., Johnson, S., ... & Schweizer, E. (1999). The researcher's own therapy allegiances: A "wild card" in comparisons of treatment efficacy. *Clinical Psychology: Science and Practice*, *6*(1), 95–106. <a href="https://doi.org/10.1093/clipsy.6.1.95">https://doi.org/10.1093/clipsy.6.1.95</a>
- Luppa, M., Heinrich, S., Angermeyer, M. C., König, H.-H., & Riedel-Heller, S. G. (2007). Cost-of-illness studies of depression. *Journal of Affective Disorders*, *98*(1–2), 29–43. https://doi.org/10.1016/j.jad.2006.07.017
- Margraf, J., Cwik, J. C., von Brachel, R., Suppiger, A., & Schneider, S. (2021). *DIPS Open Access* 1.2: Diagnostisches Interview bei psychischen Störungen. Ruhr-Universität Bochum (RUB). https://doi.org/10.46586/rub.172.149
- Martell, C. R., Dimidjian, S., Hermann-Dunn, R., Winter, L., & Lewinsohn, P. M. (2015). Verhaltensaktivierung bei Depression: Eine Methode zur Behandlung von Depression (1. Aufl). Kohlhammer.
- McCullough, J. P., Schramm, E., Penberthy, K. (2014). *CBASP as a Distinctive Treatment for Persistent Depressive Disorder*. Routledge. <a href="https://doi.org/10.4324/9781315743196">https://doi.org/10.4324/9781315743196</a>
- Menke, A., & Binder, E. B. (2014). Epigenetic alterations in depression and antidepressant treatment. *Dialoges in Clinical Neuroscience*, *16*(3), 395–404. https://doi.org/10.1159/000491431
- Michalak, J., Schultze, M., Heidenreich, T., & Schramm, E. (2015). A randomized controlled trial on the efficacy of mindfulness-based cognitive therapy and a group version of cognitive behavioral analysis system of psychotherapy for chronically depressed patients.

- Journal of Consulting and Clinical Psychology, 83(5), 951–963. https://doi.org/10.1037/ccp0000042
- Middleton, H., Shaw, I., Hull, S., & Feder, G. (2005). NICE guidelines for the management of depression. *BMJ*, 330(7486), 267–268. <a href="https://doi.org/10.1136/bmj.330.7486.267">https://doi.org/10.1136/bmj.330.7486.267</a>
- Montgomery, S. A., & Åsberg, M. (1979). A New Depression Scale Designed to be Sensitive to Change. *British Journal of Psychiatry*, *134*(4), 382–389. https://doi.org/10.1192/bjp.134.4.382
- Munder, T., Bruetsch, O., Leonhart, R., Gerger, H., & Barth, J. (2013). Researcher allegiance in psychotherapy outcome research: an overview of reviews. *Clinical Psychology Review,* 33(4), 501–511. <a href="https://doi.org/10.1016/j.cpr.2013.02.002">https://doi.org/10.1016/j.cpr.2013.02.002</a>
- Murphy, J. A., & Byrne, G. J. (2012). Prevalence and correlates of the proposed DSM-5 diagnosis of Chronic Depressive Disorder. *Journal of Affective Disorders*, 139(2), 172–180. https://doi.org/10.1016/j.jad.2012.01.033
- Murphy, J. A., Sarris, J., & Byrne, G. J. (2017). A Review of the Conceptualisation and Risk Factors Associated with Treatment-Resistant Depression. *Depression Research and Treatment*, 2017, 1–10. https://doi.org/10.1155/2017/4176825
- Nagy, G. A. et al. Reward network modulation as a mechanism of change in behavioral activation. *Behavior modification* 44, 186-213 (2020). https://doi.org/10.1177%2F0145445518805682
- Negt, P., Brakemeier, E.-L., Michalak, J., Winter, L., Bleich, S., & Kahl, K. G. (2016). The treatment of chronic depression with cognitive behavioral analysis system of psychotherapy: A systematic review and meta-analysis of randomized-controlled clinical trials. *Brain and Behavior*, *6*(8), e00486. <a href="https://doi.org/10.1002/brb3.486">https://doi.org/10.1002/brb3.486</a>
- Nemeroff, C. B., Heim, C. M., Thase, M. E., Klein, D. N., Rush, A. J., Schatzberg, A. F., Ninan, P. T., McCullough, J. P., Weiss, P. M., Dunner, D. L., Rothbaum, B. O., Kornstein, S., Keitner, G., & Keller, M. B. (2003). Differential responses to psychotherapy versus pharmacotherapy in patients with chronic forms of major depression and childhood trauma. *Proceedings of the National Academy of Sciences*, *100*(24), 14293–14296. <a href="https://doi.org/10.1073/pnas.2336126100">https://doi.org/10.1073/pnas.2336126100</a>
- Niv, Y. et al. Tonic dopamine: opportunity costs and the control of response vigor. *Psychopharmacology (Berl)* (2007). <a href="https://doi.org/10.1007/s00213-006-0502-4">https://doi.org/10.1007/s00213-006-0502-4</a>
- Norcross, J. C., & Wampold, B. E. (2011). Evidence-based therapy relationships: Research conclusions and clinical practices. *Psychotherapy*, *48*(1), 98–102. https://doi.org/10.1037/a0022161
- Reinhard, M.A., Zentz, K., Nenov-Matt, T., Barton, B.B., V. Rek, S., Goerigk, S., **Brakemeier**, **E.L.**, Musil, R., Jobst, A., Padberg, F. (accepted). Cognitive Behavioral Analysis System of Psychotherapy reduces loneliness in patients with persistent depressive disorder. *Journal of Affective Disorders Reports*
- Richards, D. A., Ekers, D., McMillan, D., Taylor, R. S., Byford, S., Warren, F. C., Barrett, B., Farrand, P. A., Gilbody, S., Kuyken, W., O'Mahen, H., Watkins, E. R., Wright, K. A., Hollon, S. D., Reed, N., Rhodes, S., Fletcher, E., & Finning, K. (2016). Cost and Outcome of Behavioural Activation versus Cognitive Behavioural Therapy for Depression (COBRA): A randomised, controlled, non-inferiority trial. *The Lancet*, *388*(10047), 871–880. https://doi.org/10.1016/S0140-6736(16)31140-0
- Robinson, L. A., Berman, J. S., & Neimeyer, R. A. (1990). Psychotherapy for the treatment of depression: a comprehensive review of controlled outcome research. *Psychological Bulletin*, 108(1), 30. <a href="https://doi.org/10.1037/0033-2909.108.1.30">https://doi.org/10.1037/0033-2909.108.1.30</a>

- Rosenbaum, S., Sherrington, C., & Tiedemann, A. (2015). Exercise augmentation compared with usual care for post-traumatic stress disorder: A randomized controlled trial. *Acta Psychiatrica Scandinavica*, *131*(5), 350–359. <a href="https://doi.org/10.1111/acps.12371">https://doi.org/10.1111/acps.12371</a>
- Russell, D. W. (1996). UCLA Loneliness Scale (Version 3): Reliability, validity, and factor structure. *Journal of personality assessment*, *66*(1), 20–40. https://doi.org/10.1207/s15327752jpa6601 2
- Rush, A. J., Carmody, T., & Reimitz, P.-E. (2000). The Inventory of Depressive Symptomatology (IDS): Clinician (IDS-C) and Self-Report (IDS-SR) ratings of depressive symptoms. *International Journal of Methods in Psychiatric Research*, *9*(2), 45–59. <a href="https://doi.org/10.1002/mpr.79">https://doi.org/10.1002/mpr.79</a>
- Sabaß, L., Padberg, F., Normann, C., Engel, V., Konrad, C., Helmle, K., Jobst, A., Worlitz, A., & Brakemeier, E.-L. (2018). Cognitive Behavioral Analysis System of Psychotherapy as group psychotherapy for chronically depressed inpatients: A naturalistic multicenter feasibility trial. *European Archives of Psychiatry and Clinical Neuroscience*, 268(8), 783–796. <a href="https://doi.org/10.1007/s00406-017-0843-5">https://doi.org/10.1007/s00406-017-0843-5</a>
- Sackeim, H. A., Aaronson, S. T., Bunker, M. T., et al. (2019). The assessment of resistance to antidepressant treatment: Rationale for the Antidepressant Treatment History Form: Short Form (ATHF-SF). *Journal of Psychiatry Research*, 113, 125–136. https://doi:10.1016/j.jpsychires.2019.03.021
- Schefft, C., Guhn, A., Brakemeier, E.-L., Sterzer, P., & Köhler, S. (2019). Efficacy of inpatient psychotherapy for major depressive disorder: a meta-analysis of controlled trials. *Acta Psychiatrica Scandinavica*, 139(4), 322–335. https://doi.org/10.1111/acps.12995
- Schramm, E., Kriston, L., Zobel, I., Bailer, J., Wambach, K., Backenstrass, M., Klein, J. P., Schoepf, D., Schnell, K., Gumz, A., Bausch, P., Fangmeier, T., Meister, R., Berger, M., Hautzinger, M., & Härter, M. (2017). Effect of Disorder-Specific vs Nonspecific Psychotherapy for Chronic Depression: A Randomized Clinical Trial. *JAMA Psychiatry*, 74(3), 233. <a href="https://doi.org/10.1001/jamapsychiatry.2016.3880">https://doi.org/10.1001/jamapsychiatry.2016.3880</a>
- Schramm, E., Schneider, D., Zobel, I., van Calker, D., Dykierek, P., Kech, S., Härter, M., & Berger, M. (2008). Efficacy of Interpersonal Psychotherapy plus pharmacotherapy in chronically depressed inpatients. *Journal of Affective Disorders*, *109*(1–2), 65–73. <a href="https://doi.org/10.1016/j.jad.2007.10.013">https://doi.org/10.1016/j.jad.2007.10.013</a>
- Schramm, E., van Calker, D., Dykierek, P., Lieb, K., Kech, S., Zobel, I., Leonhart, R., & Berger, M. (2007). An Intensive Treatment Program of Interpersonal Psychotherapy Plus Pharmacotherapy for Depressed Inpatients: Acute and Long-Term Results. *American Journal of Psychiatry*, 164(5), 768–777. https://doi.org/10.1176/ajp.2007.164.5.768
- Schramm, E., Zobel, I., Dykierek, P., Kech, S., Brakemeier, E.-L., Külz, A., & Berger, M. (2011). Cognitive behavioral analysis system of psychotherapy versus interpersonal psychotherapy for early-onset chronic depression: A randomized pilot study. *Journal of Affective Disorders*, 129(1–3), 109–116. https://doi.org/10.1016/j.jad.2010.08.003
- Schramm, E., Zobel, I., Schoepf, D., Fangmeier, T., Schnell, K., Walter, H., Drost, S., Schmidt, P., Brakemeier, E.-L., Berger, M., & Normann, C. (2015). Cognitive Behavioral Analysis System of Psychotherapy versus Escitalopram in Chronic Major Depression. *Psychotherapy and Psychosomatics*, 84(4), 227–240. https://doi.org/10.1159/000381957
- Schwarzer, R., & Jerusalem, M. (1995). Generalized Self-Efficacy scale. In J. Weinman, S. Wright, & M. Johnston, Measures in health psychology: A user's portfolio. Causal and control beliefs (pp. 35-37). Windsor, UK: NFER-NELSON.

- Seidl, H., Bowles, D., Bock, J.-O., Brettschneider, C., Greiner, W., König, H.-H., & Holle, R. (2014). FIMA Fragebogen zur Erhebung von Gesundheitsleistungen im Alter: Entwicklung und Pilotstudie. *Das Gesundheitswesen*, 77(01), 46–52. https://doi.org/10.1055/s-0034-1372618
- Shinohara, K., Honyashiki, M., Imai, H., Hunot, V., Caldwell, D. M., Davies, P., Moore, T. H., Furukawa, T. A., & Churchill, R. (2013). Behavioural therapies versus other psychological therapies for depression. *Cochrane Database of Systematic Reviews*. https://doi.org/10.1002/14651858.CD008696.pub2
- Smith, B. W., Dalen, J., Wiggins, K., Tooley, E., Christopher, P., & Bernard, J. (2008). The brief resilience scale: assessing the ability to bounce back. *International journal of behavioral medicine*, *15*(3), 194-200. https://doi.org/10.1080/10705500802222972
- Snarski, M., Scogin, F., DiNapoli, E., Presnell, A., McAlpine, J., & Marcinak, J. (2011). The Effects of Behavioral Activation Therapy With Inpatient Geriatric Psychiatry Patients. *Behavior Therapy*, 42(1), 100–108. <a href="https://doi.org/10.1016/j.beth.2010.05.001">https://doi.org/10.1016/j.beth.2010.05.001</a>
- Spates, C. R., Pagoto, S. L., & Kalata, A. (2006). A qualitative and quantitative review of behavioral activation treatment of major depressive disorder. *The Behavior Analyst Today*, 7(4), 508–521. https://doi.org/10.1037/h0100089
- Staebler, K., Helbing, E., Rosenbach, C., & Renneberg, B. (2011). Rejection sensitivity and borderline personality disorder. *Clinical psychology & psychotherapy*, *18*(4), 275–283. https://doi.org/10.1002/cpp.705
- Tadić, A., Müller-Engling, L., Schlicht, K. F., Kotsiari, A., Dreimüller, N., Kleimann, A., Bleich, S., Lieb, K., & Frieling, H. (2014). Methylation of the promoter of brain-derived neurotrophic factor exon IV and antidepressant response in major depression. *Molecular Psychiatry*, 19(3), 281–283. <a href="https://doi.org/10.1038/mp.2013.58">https://doi.org/10.1038/mp.2013.58</a>
- Vinkers, C. H., Geuze, E., van Rooij, S. J. H., Kennis, M., Schür, R. R., Nispeling, D. M., Smith, A. K., Nievergelt, C. M., Uddin, M., Rutten, B. P. F., Vermetten, E., & Boks, M. P. (2021). Successful treatment of post-traumatic stress disorder reverses DNA methylation marks. *Molecular Psychiatry*, 26(4), 1264–1271. https://doi.org/10.1038/s41380-019-0549-3
- Wagner, T., Fydrich, T., Stiglmayr, C., Marschall, P., Salize, H-J., Renneberg, B., Fleßa, S., & Roepke, S. (2014). Societal cost-of-illness in patients with borderline personality disorder one year before, during and after dialectical behavior therapy in routine outpatient care. Behaviour Research and Therapy, 61, 12–22. <a href="https://doi.org/10.1016/j.brat.2014.07.004">https://doi.org/10.1016/j.brat.2014.07.004</a>
- Weck, F., Hautzinger, M., Heidenreich, T., & Stangier, U. (2010). Erfassung psychotherapeutischer Kompetenzen: Validierung einer deutschsprachigen Version der Cognitive Therapy Scale. *Zeitschrift für Klinische Psychologie und Psychotherapie*, *39*(4), 244–250. <a href="https://doi.org/10.1026/1616-3443/a000055">https://doi.org/10.1026/1616-3443/a000055</a>
- Wiersma, J. E., Van Schaik, D. J. F., Hoogendorn, A. W., Dekker, J. J., Van, H. L., Schoevers, R. A., Blom, M. B. J., Maas, K., Smit, J. H., McCullough Jr., J. P., Beekman, A. T. F., & Van Oppen, P. (2014). The Effectiveness of the Cognitive Behavioral Analysis System of Psychotherapy for Chronic Depression: A Randomized Controlled Trial. *Psychotherapy and Psychosomatics*, 83(5), 263–269. <a href="https://doi.org/10.1159/000360795">https://doi.org/10.1159/000360795</a>
- Wingenfeld, K., Spitzer, C., Mensebach, C., Grabe, H.J., Hill, A., Gast, U., Schlosser, N., Höpp, H., Beblo, T., Driessen, M., 2010. The German Version of the Childhood\_Trauma Questionnaire (CTQ): Preliminary Psychometric Properties. *PPmP: Psychotherapie Psychosomatik Medizinische Psycholologie, 60*, 442–450. <a href="https://doi.org/10.1055/s-0030-1247564">https://doi.org/10.1055/s-0030-1247564</a>

- Williams, J. B. (1988). A structured interview guide for the Hamilton Depression Rating Scale. *Archives of General Psychiatry*, 45(8), 742–747.
- Wilmers, F., Munder, T., Leonhart, R., Herzog, T., Plassmann, R., Barth, J., & Linster, H. W. (2008). Die deutschsprachige Version des Working Alliance Inventory Short revised (WAI-SR) Ein schulenübergreifendes, ökonomisches und empirisch validiertes Instrument zur Erfassung der therapeutischen Allianz. *Klinische Diagnostik und Evaluation* (1. Aufl.), Vandenhoeck & Ruprecht GmbH.
- Zheleznyakova, G. Y., Cao, H., & Schiöth, H. B. (2016). BDNF DNA methylation changes as a biomarker of psychiatric disorders: Literature review and open access database analysis. *Behavioral and Brain Functions.*
- Zimmermann, J., Woods, W. C., Ritter, S., Happel, M., Masuhr, O., Jaeger, U., Spitzer, C., & Wright, A. (2019). Integrating structure and dynamics in personality assessment: First steps toward the development and validation of a personality dynamics diary. *Psychological assessment*, *31*(4), 516–531. <a href="https://doi.org/10.1037/pas0000625">https://doi.org/10.1037/pas0000625</a>